#### GlaxoSmithKline group of companies

**Division:** World Wide Development **Retention Category:** GRS019

Information Type: Reporting and Analysis Plan

**Title:** Reporting and Analysis Plan for AMB112529:

A randomized, open label study comparing safety and efficacy parameters for a high and a low dose of ambrisentan (adjusted for body weight) for the treatment of pulmonary arterial

hypertension in paediatric patients aged 8 years up to 18 years.

**Compound Number:** GSK1325760

Effective Date: 22-MAY-2018

**Description**: This document outlines the safety and efficacy reporting planned for protocol AMB112529 by GlaxoSmithKline (GSK).

**Identifier/Version Number:** Version 1.0

**Subject:** GSK1325760, Pulmonary Artery Hypertension; Reporting; Tables, Figures, Listings (TFLs)

Author's Name, Title and Functional Area: PPD Managing Director, Hartington Statistics and Data Management Ltd.

#### Approved by:

PPD Date

Director,

Clinical Statistics 22-MAY-2018

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| AB | BREVIA | ATIONS | | | 5 |
| 1. | INTRO | DUCTIO | N | | 7 |
| 2. | STUD | Y OBJEC | TIVE(S) AN | D ENDPOINT(S) | 7 |
| | 2.1. | | | 2 2 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 | |
| | | 2.1.1. | | bjective | |
| | | 2.1.2. | Secondary | Objectives | 7 |
| | 2.2. | • | | | |
| | | 2.2.1. | | ndpoints | |
| | | 2.2.2. | | / Endpoints | |
| | | | 2.2.2.1.<br>2.2.2.2. | Pharmacokinetics | |
| | | | | Efficacy Exploratory | |
| | | | 2.2.2.4. | Other | |
| | 2.3. | Statistica | | es | |
| | 2.4. | | | K) and PK/Pharmacodynamic (PD) hypotheses | |
| 3. | STUD | Y DESIG | N | | 8 |
| 0. | 3.1. | | | | |
| | D. 44. | | 11/050 | | • |
| 4. | | | | | |
| | 4.1.<br>4.2. | | • | | |
| | 4.2. | 4.2.1. | • | n the conduct of the study or planned analyses | |
| 5. | SAMP | LE SIZE | CONSIDER | ATIONS | 10 |
| 6. | ΛΝΑΙ | veie bot | DI II ATIONS | | 10 |
| 0. | ANAL | 1313 PU | POLATIONS | · | 10 |
| 7. | TREA | | | DNS | |
| | 7.1. | Data Dis | splay Treatm | nent and Other Sub-group Descriptors | 10 |
| 8. | GENE | RAL CON | NSIDERATIO | ONS FOR DATA ANALYSES | 10 |
| | 8.1. | Examina | ation of Subg | groups | 10 |
| _ | | | | VITION 6 | |
| 9. | | | | NTIONS | |
| | 9.1. | 9.1.1. | | val and Missing Data | |
| | | 9.1.1. | | ficacy Outcomes Data<br>E data | |
| | | 9.1.2. | | ates (other than for AEs) | |
| | | 9.1.4. | | ems on SF-10 | |
| | 9.2. | - | | ormed Data | |
| | | 9.2.1. | | | 12 |
| | | 9.2.2. | | om baseline and percentage change from | |
| | | 9.2.3. | | change from baseline categorisation 1 | |
| | | 9.2.4. | | class change from baseline categorisation 2 | |
| | | 9.2.5. | Study Day | | 13 |

| | 9.3.<br>9.4. | | Age Calculation Duration of Exposure Transformations for Efficacy Outcomes Treatment Compliance Rates ent Windows f Clinical Concern Laboratory Parameters Vital Signs | 14<br>14<br>15<br>15 |
|---|---|---|---|---|
| 10. | STUDY<br>10.1.<br>10.2.<br>10.3.<br>10.4.<br>10.5.<br>10.6.<br>10.7. | Disposition<br>Protocol<br>Demogration<br>Medical (Prior and<br>Treatment | ATION | 17<br>17<br>18<br>18 |
| 11. | SAFET<br>11.1.<br>11.2.<br>11.3. | Extent of<br>Adverse<br>Adverse<br>Product a | SES Exposure Events Events Leading to Discontinuation of Investigational and/or Withdrawal from the Study and Other Significant Events | 19<br>19 |
| | 11.11.<br>11.12. | Deaths a<br>Adverse<br>Non-seric<br>Clinical L<br>Liver Eve<br>Vital Sign<br>Physical<br>12-Lead<br>Endocrin | Events of Special Interest Dus Adverse Events Baboratory Evaluations Examination ECG Ology Cies (as applicable) | 20<br>21<br>21<br>21<br>21<br>21 |
| 12. | 12.1. | Explorate | LYSESalysesalyses | 23 |
| 13. | 13.1.<br>13.2. | Pharmac<br>Pharmac | RMACOLOGY DATA ANALYSES<br>cokinetic Analysescodynamic Analysescokinetic/Pharmacodynamic Analyses | 23 |
| 14. | BIOMA | RKER D | ATA ANALYSIS | 23 |
| 15. | PHARI | MACOGE | NETIC DATA ANALYSES | 23 |
| 16. | VIRAL | GENOTY | PING/PHENOTYPING | 24 |
| 17. | REFER | RENCES. | | 24 |
| 18 | ΑΤΤΔΟ | HMENTS | | 25 |

| | 18.1. | Table of Contents for Data Display Specifications | 25 |
|-----|-------|---------------------------------------------------|-----|
| | | 18.1.1. Tables | |
| | | 18.1.2. Listings | 31 |
| | | 18.1.3. Figures | |
| | 18.2. | Data Display Specifications | |
| 19. | APPE | ENDICES | 145 |
| | 19.1. | Appendix 1 – IDSL Age Calculation | 145 |

#### **ABBREVIATIONS**

AE adverse event

ALT alanine aminotransferase
AST aspartate aminotransferase

ATC Anatomical Therapeutic Chemical

DBF Database Freeze

eCRF Electronic case report form

ECG electrocardiogram
GSK GlaxoSmithKline

IDMC Independent Data Monitoring Committee

IP Investigational product

ITT Intent-to-Treat

MedDRA Medical Dictionary for Regulatory Activities

6MWD 6 minute walking distance

NT-Pro BNP N-terminal pro-B-type natriuretic peptide

PAH pulmonary arterial hypertension

PD pharmacodynamic
PK pharmacokinetic
PT Preferred Term
RA Right Atrial

RAP Reporting and Analysis Plan

RUCAM Roussel Uclaf Causality Assessment Method

RV Right Ventricular

SAE Serious Adverse Event

SAS Statistical Analysis System

SD Standard deviation
SOC System Organ Class

TAPSE Tricuspid Annular Plane Systolic Excursion

TFLs Tables, Figures, Listings
TRJ Tricuspid Regurgitant Jet
WHO World Health Organization

## **Trademark Information**

| Trademarks of the GlaxoSmithKline group of companies |
|------------------------------------------------------|
| AMBRISENTAN |
| FLOLAN |

| GlaxoSmithKline group of companies |
|------------------------------------|
| Adcirca |
| C RIBA |
| Letairis |
| NONMEM |
| Remodulin |
| Revatio |
| Thelin |
| Tracleer |
| Ventavis |
| Viagra |

#### 1. INTRODUCTION

This Reporting and Analysis Plan (RAP) outlines the safety and efficacy reporting planned for protocol AMB112529 for provision to GSK.

In this RAP, reference is made to the protocol AMB112529 dated 2<sup>nd</sup> February 2011, and subsequent amendments.

## 2. STUDY OBJECTIVE(S) AND ENDPOINT(S)

## 2.1. Study Objective(s)

## 2.1.1. Primary Objective

The primary objective is the safety and tolerability of ambrisentan in the paediatric pulmonary arterial hypertension (PAH) population.

## 2.1.2. Secondary Objectives

The secondary objectives are the pharmacokinetics and efficacy of ambrisentan in the paediatric pulmonary arterial hypertension (PAH) population.

## 2.2. Study Endpoint(s)

## 2.2.1. Primary Endpoints

- Adverse Events.
- Serious Adverse Events.
- Clinical laboratory parameters.
- Physical examination
- Vital Signs.
- Pubertal development (change from baseline in endocrinology assessments at Weeks12 and 24).

## 2.2.2. Secondary Endpoints

#### 2.2.2.1. Pharmacokinetics

- Population pharmacokinetic assessment based on one plasma sample per subject at Weeks 4 (trough), 8 (0.5 to 4 hours post-dose), 12 (trough), 16 (0.5 to 4 hours postdose), 20 (4 to 22 hours post-dose), and 24 (trough).
- Pharmacokinetic/pharmacodynamic modelling.

#### 2.2.2.2. Efficacy

- The change from baseline in the 6 minute walking distance (6MWD) test evaluated after 24 weeks of therapy.
- Mean changes from baseline in the 6MWD test at Weeks 4, 8, 12, 16, and 20.
- The time to clinical worsening of PAH.

- The change from baseline in Subject Global Assessment to Week 24 using the SF-10 health survey for children.
- The change from baseline in World Health Organization (WHO) functional class to Week 24.
- Change from baseline in plasma N-Terminal pro-B-type Natriuretic Peptide (NT-Pro BNP) concentration at Week 24.
- School days missed due to PAH. (Note that this is not defined as an efficacy endpoint in the protocol but has been added to the RAP.)

#### 2.2.2.3. Exploratory

■ The change from baseline in major prognostic factors based on echocardiogram: pericardial effusion, right atrial (RA) pressure, tricuspid annular plane systolic excursion (TAPSE), eccentricity index (systolic and diastolic), and right ventricular (RV) pressure by tricuspid regurgitant jet (TRJ) velocity to Week 24.

#### 2.2.2.4. Other

Change from baseline in cardiopulmonary hemodynamics at Week 24 (a substudy in subjects enrolled at centres where the collection of hemodynamic data is considered part of the standard of care).

#### 2.3. Statistical Hypotheses

No formal hypothesis is planned.

## 2.4. Pharmacokinetic (PK) and PK/Pharmacodynamic (PD) hypotheses

Any statistical hypothesis relating to the pharmacokinetic endpoints will be described in a separate RAP. The analysis will be the responsibility of the Department of Clinical Pharmacology Modeling and Simulation (CPMS), Quantitative Sciences, GSK.

#### 3. STUDY DESIGN

This study is a 6-month (24-week), randomized, open label evaluation of the safety, tolerability and efficacy of a high and low dose ambrisentan (adjusted for body weight) in 66 subjects (33 per treatment group) aged 8 years up to 18 years with PAH. The study will include a screening/baseline period and a treatment period. The treatment period will be 24 weeks or until the subject's clinical condition deteriorates to the point that alternative/additional treatment is necessary. Subjects who participate in the study will be eligible to enrol into study AMB 114588.

For further details regarding the study design, please refer to the protocol.

#### 3.1. Randomisation

All subjects who meet the inclusion and exclusion criteria will be randomized to one of two dose groups (Low dose or High dose, based on body weight) of ambrisentan according to a computer-generated randomisation schedule.

| Body Weight | Low Dose | High Dose |
|-----------------|----------|-----------|
| >=50kg | 5 mg | 10 mg |
| >=35 and <50 kg | 5 mg | 7.5 mg |
| >=20 and <35 kg | 2.5 mg | 5 mg |

To ensure balance with respect to the number of patients assigned to each treatment group, the allocation schedule will be generated in blocks. Each subject will be assigned to a pack number according to the predefined randomisation list. A central Interactive Voice Response System (IVRS) will be used for treatment assignment.

Randomization will be stratified by the age groups 8 years up to 11 years and 12 years up to 18 years and by aetiology of PAH as follows:-

- idiopathic;
- heritable [familial];
- secondary to connective tissue disease; and
- persistent despite surgical repair of atrial septal defects, ventricular septal defects, atrio-ventricular septal defects, and persistent patent ductus.

Subjects will be assigned to study treatment in accordance with the randomization schedule.

#### 4. PLANNED ANALYSES

## 4.1. Interim Analyses

The interim analyses conducted by the Independent Data Monitoring Committee (IDMC) are planned for this study. These analyses are described in a dedicated IDMC RAP.

To facilitate the communication between GSK and regulatory agency, an interim analysis was added post the finalization of the study protocol. For data collected up until January 2018, all safety, tolerability, pharmacokinetics and efficacy data will be reviewed, analysed and summarised.

## 4.2. Final Analysis

This analysis plan outlines the final analysis that will be performed on the safety and efficacy endpoints of this study, once Database Freeze (DBF) has taken place.

## 4.2.1. Changes in the conduct of the study or planned analyses

The final analyses were as planned in the protocol except for the following:-

- Protocol, Section 8.3.5.4 states summary analysis of the differences between Low and High groups will be performed. However, due to low subject numbers, this is not presented in this RAP.
- School days missed due to PAH has been added to the RAP.

#### 5. SAMPLE SIZE CONSIDERATIONS

Due to the low prevalence of the disease in children, sample size was based on feasibility rather than formal power calculations. Recruitment of approximately 66 subjects (33 per treatment group with no prespecified number in each age group/aetiology stratum) is felt to be achievable within a reasonable period of time (~ 2 years) minimizing any impact of changing practice on the conduct and interpretation of the study.

#### 6. ANALYSIS POPULATIONS

The Intent-to-Treat (ITT) Population will consist of all randomized subjects who received at least 1 dose of study drug. For the ITT population, subjects were considered as belonging to their randomized treatment group, regardless of the actual dose of ambrisentan received. The ITT population will be used in all efficacy summaries.

The Safety Population is defined as all randomized subjects who received at least 1 dose of study drug. Subjects were considered as belonging to the treatment group according to highest dose received. The safety population will be used in all safety summaries.

#### 7. TREATMENT COMPARISONS

Treatment comparisons will be between low dose and high dose ambrisentan, by way of summary tables, figures and listings.

#### 7.1. Data Display Treatment and Other Sub-group Descriptors

In the study report data displays, the treatment group descriptors will be the following:

- Ambrisentan Low Dose
- Ambrisentan High Dose

#### 8. GENERAL CONSIDERATIONS FOR DATA ANALYSES

All programming of tables, figures and listings will be performed using Statistical Analysis System (SAS) version 8.2 or higher.

## 8.1. Examination of Subgroups

Selected safety and efficacy outputs will be produced by age strata (8-11, 12-18 years).

Selected outputs will also be produced for patients enrolled at centres in Japan to support registration activities.

#### 9. DATA HANDLING CONVENTIONS

All data displays will be presented according to the GSK's Integrated Data Standards Library (IDSL) statistical display principles. The file extension used for landscape tables and listings will be L10, with point size of 10, line size of 108 and 43 lines per page.

Where data are sparse, empty tables may be produced with the "Data too sparse for table to be produced" or "No Data to Report" or similar.

All data collected on the electronic case report form (eCRF) will be listed. Data collected outside of the eCRFs (eg. labs, SF10) will also be listed. All listings will be presented by treatment group, centre identification and subject identification number.

#### 9.1. Premature Withdrawal and Missing Data

Subjects who withdraw from the study prior to Week 24 will not be replaced and all information obtained from them will be included in the summaries.

#### 9.1.1. Missing Efficacy Outcomes Data

No imputation will be made for any missing numerical data, unless otherwise specified.

Missing data will generally not be considered in the calculation of percentages (i.e., the denominator will not include subjects who have missing data at a given time point).

#### 9.1.2. Missing AE data

Where a start date for an adverse event (AE) is partial or missing, the following imputation rules will be applied:

- If day portion is missing, set day to 1.
- If month portion is missing, set month to January.
- If the date is completely missing, or if the date imputed using the above rules is prior to the first dose date, set the date to first dose date.

Where an end date for an AE is partial or missing, the following imputation rules will be applied. These will only be applied to AEs that are resolved; if they are not resolved then nothing will be imputed.

- If day portion is missing, set day to the last day of the month.
- If month portion is missing, set month to December.
- If the date is completely missing, or if the date imputed using the above rules is after the treatment end date, set the date to the treatment end date or if the treatment end date is missing then set to date of discontinuation.

No further imputation will be performed for missing data.

#### 9.1.3. Missing Dates (other than for AEs)

For any data type that collects partial dates, impute missing day as 01 and missing month as January. If date is completely missing then date should remain missing.

Where the start date of study medication is missing, the date of randomisation will be used. Where end date of study medication is partial or missing, the last complete non-missing date of dosing will be used as the last date for determining duration of exposure.

#### 9.1.4. Missing Items on SF-10

The SF-10 will be scored in accordance with the developer's guidelines. Out-of-range values are converted to missing values and no algorithm is used to estimate missing values. The Physical and Psychosocial summary scores are not calculated if any component scores are missing.

#### 9.2. Derived and Transformed Data

All listings will include all subjects that have the relevant data for each listing.

The number of subjects (N) in each treatment group and overall for the population being summarised, will be displayed in each table unless specified otherwise.

For continuous data, the following summary statistics will be presented: n, mean, standard deviation (SD), median, upper and lower quartiles, minimum and maximum.

Mean and median values will be reported to one decimal place greater than the original data they were collected from while the SD will be reported to two decimal places greater than the original data however, if this results in a value of 0.00 being presented then a zero (0) will be presented. Minimum and maximum values will be reported with the same precision as they were collected.

All text fields must be left justified. Numeric or numeric with some text specification (e.g., not done, unknown, <4.5, ...) must be right justified.

The format for dates will be DDMMMYYYY.

All tables and listings will have the protocol number and population in the top left-hand corner and the page number in the form of page x of n will be presented in the top right-hand corner. In the bottom left-hand corner of tables and listings the name of the person who created the output followed by a colon, the output filepath and the date and time of the production of the output, in the form DDMMMYYYY HH:MM, will be displayed.

If a count in a table summary is zero (0) then a percentage will not be presented.

To determine whether an adverse event is on-treatment and a medication is prior or concomitant, imputation of missing or partial start and stop dates is required (see RAP Section 9.1.2 and Section 9.1.3). Imputed dates will not be listed and adverse event duration will not be calculated if the start date or stop date had to be imputed.

#### 9.2.1. Baseline

Baseline values are those collected prior to the first dose. Therefore if a subject has no data for a parameter on Day 1 (prior to first dose) then the data from their last pretreatment assessment will be used.

#### 9.2.2. Change from baseline and percentage change from baseline

For untransformed data change from baseline at Week X will be calculated as Week X value minus baseline value. The percentage change from baseline at Week X will be calculated as:  $100 \times (\text{Week X value} - \text{baseline value}) / \text{baseline value}$ .

For log-transformed data (see Section 9.2.8), ratio to baseline expressed as percentage change will be calculated by taking the mean change on the log scale, exponentiating, subtracting 1 and multiplying by 100.

(Exp(mean of (Log x - Log baseline)) -1)\*100

#### 9.2.3. WHO FC change from baseline categorisation 1

Note that based on the study inclusion criteria subjects must have a WHO FC of II or III at baseline. Change from baseline at Week X will be calculated as Week X value minus baseline value, thus categories may be -2, -1, 0, +1, +2.

| | | | Post Baseline WHO FC | | |
|--------------|----|----|----------------------|-----|----|
| | | I | П | III | IV |
| Baseline WHO | II | -1 | 0 | +1 | +2 |
| FC | Ш | -2 | -1 | 0 | +1 |

#### 9.2.4. WHO FC class change from baseline categorisation 2

Improved = -1 or -2 in Change from Baseline Categorisation No change = 0 in Change from Baseline Categorisation Deteriorated = +1 or +2 in Change from Baseline Categorisation

#### 9.2.5. Study Day

Study Day 1 is defined as the day of the first dose of study drug.

**Relative Day to start of study medication** for an Event is defined as:

Date of event - Date of first study medication + 1, if the event is on or after the first dose date.

Date of event - Date of first study medication, if the event is prior to the first dose date.

#### **Relative Day to end of medication** for an Event is defined as:

Date of event - Date of last study medication +1, if the event is on or after the last dose date.

Date of event - Date of last study medication, if the event is prior to the last dose date.

#### 9.2.6. Age Calculation

Age in years at baseline will be derived as a whole number according to the IDSL standard algorithm (see Appendix 1).

#### 9.2.7. Duration of Exposure

Duration of exposure to study drug will be calculated in days as (Treatment stop date – Treatment start date) + 1.

#### 9.2.8. Transformations for Efficacy Outcomes

A log transformation will be applied to NT-proBNP data.

Summaries of the relative changes from baseline based on analysis of log-transformed data will include the geometric mean and coefficient of variation (calculated as below based on the logged values) and the geometric mean of the ratio of the value of the endpoint at the time point of interest to the baseline value (see Section 9.2.2).

Geometric mean =  $\exp(\mu)$ 

Coefficient of variation =  $100 \text{ x} \sqrt{\left[\exp(\sigma^2) - 1\right]}$ 

#### 9.2.9. Treatment Compliance Rates

Compliance to study medication is recorded at each visit in one of the following categorical groups:-

- 0% compliant (subject did not take any doses)
- >0% and < 80% compliant (subject missed a number of doses)
- >=80% and <=120%, (number of doses taken was within compliance range)
- >120% compliant (number of doses taken exceeds compliance limits)

At the subject level compliance rate is calculated as

100\*(the number of visits at which the subject was compliant (i.e.  $\geq$ 80% and  $\leq$ 120%) / (the sum of all study visits for the subject).

At a treatment group level compliance rate is calculated as

100\*(the total number of visits at which all subjects in that group were compliant (i.e.  $\geq$  80% and  $\leq$  120%)) / (the sum of all study visits for all subjects in that group).

#### 9.3. Assessment Windows

All data will be reported for the whole study period.

Unscheduled assessments will not be slotted to a particular time point, but will remain as unscheduled unless otherwise specified.

Time points relating to nominal visits will be used in tables, figures and listings.

Time to clinical worsening of PAH and time to liver event will be calculated using the date of assessment.

## 9.4. Values of Clinical Concern

## 9.4.1. Laboratory Parameters

The following values of potential clinical concern will be considered:

| Values of potential clinical concern values will be defined for laboratory parameters as follows:Parameter | Code | Units | Low<br>Concern<br>Value (SI<br>units) | High<br>Concern<br>Value (SI<br>units) | Worse case direction |
|---|---|---|---|---|---|
| Hematology | | | | | |
| Hemoglobin | HGB | G/L | Males: < 98 Females: < 91 | Males: > 180.0<br>Females: > 161.0 | Low |
| Hematocrit | НСТ | %<br>(1) | Males:<br>< 32.0<br>(<0.32)<br>Females:<br><29.0<br>(<0.29) | Males: > 54.0 (>0.54) Females: > 50.6 (>0.506) | Low |
| Platelets | PLATE | 10^9/L<br>(same as<br>GI/L) | < 100 | > 500 | Low |
| Chemistry | | | | | |

| Values of potential clinical concern values will be defined for laboratory parameters as follows: <b>Parameter</b> | Code | Units | Low<br>Concern<br>Value (SI<br>units) | High<br>Concern<br>Value (SI<br>units) | Worse case direction |
|---|---|---|---|---|---|
| Total bilirubin | BILTOT | UMOL/<br>L | None | >= 34.2 | High |
| AST | ASAT | IU/L | None | >= 3 x<br>ULN | High |
| ALT | ALAT | IU/L | None | >= 3 x<br>ULN | High |
| GGT | GGT | IU/L | None | >= 3 x<br>ULN | High |
| Creatinine | CREAT | UMOL/<br>L | None | >= 176.8 | High |

#### 9.4.2. Vital Signs

The following criteria will be used to determine whether a subject's vital signs (blood pressure and heart rate) lie outside a pre-determined range of clinical concern:

| Parameter | Code | Units | Low Concern<br>Value | High Concern Value |
|---|---|---|---|---|
| Heart Rate | PUL | Bpm | < 50 | > 120 |
| Systolic | SYS | mm Hg | < 80 | > 160 mm Hg<br>> 30 mm Hg change from<br>Baseline |
| Diastolic | DIA | mm Hg | < 40 | > 110 mm Hg<br>> 20 mm Hg change from<br>Baseline |
| Body weight | WT | Kg | < 20 | |

#### 10. STUDY POPULATION

Study population data will be presented for the Intent-to-Treat Population unless otherwise specified.

## 10.1. Disposition of Subjects

The number of subjects eligible for each of the analysis populations will be summarised by treatment group and overall, and by country and centre.

The number of subjects completing/withdrawing from the study along with the reasons for withdrawal will be summarised by treatment group and overall.

#### 10.2. Protocol Deviations

The number of subjects with important protocol deviations will be summarised by treatment group and overall.

A summary of subjects who did not satisfy all inclusion and exclusion criteria will be provided by treatment group.

The protocol deviations will be reviewed by the clinical team after the database release and prior to the database freeze, to determine which ones are considered to be important.

## 10.3. Demographic and Baseline Characteristics

The number and percentage of subjects in each category for categorical variables or summary statistics for continuous variables will be summarised by treatment group and overall. These include age, age strata, sex, child-bearing potential, ethnicity and geographic ancestry, aetiology of PAH strata, duration of PAH, PAH therapy use, WHO FC score and 6 minute walk distance.

#### 10.4. Medical Conditions

The number and percentage of subjects with past or current medical conditions will be summarised by treatment group and overall, for any condition and by condition classification.

#### 10.5. Prior and Concomitant Medications

The GSK drug dictionary will be used to code drug names.

Prior medications are those that started and stopped prior to the date of first study treatment. Ongoing medications at baseline are those started before first dose date of study drug, which were continued during the treatment phase.

Concomitant medications are defined as:-

- Medications that start prior to or on the date of first study treatment and that stopped prior to the date of last study treatment,
- Medications that start prior to or on the date of first study treatment and continued after the date of last study treatment,
- Medications that start after the date of first study treatment and that stopped prior to the date of the last study treatment,
- Medications that start after the date of first study treatment and continued after the date of last study treatment.

Any medications that started after the last study treatment are classed as post-treatment medications.

Note that it will be assumed that the medication has been taken by the medication start and stop dates recorded in the eCRF.

The number and percentage of subjects with concomitant medications will be summarised by Anatomical Therapeutic Chemical (ATC) Classification System code and preferred term, by treatment group and overall.

The number and percentage of subjects with ongoing (at baseline) and concomitant PAH therapy at Week 24 will be summarised by preferred term, by treatment group and overall. The ATC codes from the GSKDrug dictionary for the groupings of PAH therapy will be agreed with the Clinical Safety Group and provided in a separate file. This includes:

- PDE5i
- Prostanoid

#### 10.6. Treatment Compliance

At each visit, treatment compliance will be recorded as 0%, >0% - <80%, =>80% - <=120% and >120%.

The number and percentage of subjects in each compliance category will be summarised at each visit by treatment group and overall.

#### 10.7. Long-Term Study (AMB 114588)

The number and percentage of subjects continuing in study AMB 114588 will be summarised by treatment group and overall.

#### 11. SAFETY ANALYSES

Safety data will be presented for the Safety Population unless otherwise specified.

## 11.1. Extent of Exposure

The number of days of exposure to study drug will be summarised by treatment group and overall.

This number of days of exposure will be categorised in 30 day intervals as follows: <=30 days, 31-60 days, 61-90 days etc.

The number and percentage of subjects in each of these categories will be summarised by treatment group and overall.

#### 11.2. Adverse Events

All AEs will be categorised into Preferred Term (PT) and associated System Organ Class (SOC) using the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary.

Only treatment-emergent adverse events (TEAEs) will be included in summary tables.

TEAEs are defined as those events that start on or after first dose date of study treatment.

Any subject with at least one reported TEAE will be classified as a subject with:

- A TEAE.
- A TEAE leading to study treatment discontinuation (definitive or temporary),
- A TEAE leading to study withdrawal,
- At least one serious TEAE.

The numbers and percentages of subjects with at least one reported TEAE will be summarised by treatment group and overall according to:

- PT,
- SOC and PT.
- SOC and PT by intensity,
- SOC and PT by relationship to study treatment,
- PT by action taken with investigational product (IP).

Recurring TEAEs (i.e. successive TEAEs classified with the same PT) for a given subject will only be counted once and only their most severe intensity will be tabulated.

The cumulative incidence of each TEAE will also be summarised by SOC and PT and the following categories: <2 weeks, <4 weeks, <12 weeks, <16 weeks, <20 weeks and <24 weeks.

TEAEs will be listed by SOC and PT, by treatment with the number of subjects who experienced the event and their subject numbers presented. A more detailed listing will also be produced for all subjects who experienced an AE.

# 11.3. Adverse Events Leading to Discontinuation of Investigational Product and/or Withdrawal from the Study and Other Significant Adverse Events

The numbers and percentages of subjects with at least one reported TEAE leading to discontinuation of the investigational product or withdrawal from the study will be summarised by SOC and PT for each treatment group and overall.

#### 11.4. Deaths and Serious Adverse Events

Summary tables detailed in Section 11.2 and Section 11.3 (with the exception of cumulative incidence) will be repeated for serious TEAEs.

Summary tables will also be presented for serious TEAEs by PT and outcome for each treatment group and overall.

A summary of serious TEAEs displaying the number of subjects and occurrences will also be presented.

In addition, the number of subjects with fatal TEAEs and fatal TEAEs related to IP will be summarised by SOC and PT for each treatment group and overall.

## 11.5. Adverse Events of Special Interest

Summary tables detailed in Section 11.2 and Section 11.3 (with the exception of tables by maximum intensity/grade, action taken and relation to IP) will be repeated for AEs of special interest. MedDRA preferred terms and codes for AEs of special interest will be agreed with Clinical Safety Group and provided in a separate file.

The adverse events of special interest are:

- Anaemia
- Hepatoxicity

- Hypersensitivity
- Hypotension
- Male infertility
- Oedema/fluid retention

#### 11.6. Non-serious Adverse Events

A summary of the most common (>=5%) non-serious TEAEs displaying the number of subjects and occurrences will also be presented.

#### 11.7. Clinical Laboratory Evaluations

Absolute values and changes from baseline of laboratory data will be summarised for each visit, by treatment group and overall.

Separate tables will be presented for haematology data, clinical chemistry data and endocrine data (females only).

The number and percentages of subjects with laboratory values above and below reference ranges for potential clinical concern described in Section 9.4.1 will be summarised for each visit, by treatment group and overall

#### 11.8. Liver Events

The number and percentage of subjects reporting a liver event will be summarised: overall, during and post study treatment.

The following will be listed by treatment group, for subjects with liver events:-

- liver chemistry result involved in the event.
- Time from first and last dose to start of event
- Patient specific information for liver events
- Medical conditions.
- Liver biopsy details.
- Liver imaging details.

## 11.9. Vital Signs

Absolute values and changes from baseline of vital signs data will be summarised for each visit, by treatment group and overall.

The number and percentages of subjects with vital signs values or change from baseline values above and below reference ranges for potential clinical concern described in Section 9.4.2 will be summarised for each visit, by treatment group and overall.

## 11.10. Physical Examination

Physical examination at each visit will be summarised by treatment group and overall.

#### 11.11. 12-Lead ECG

The number and percentages of subjects with electrocardiogram (ECG) abnormalities (clinically significant and not clinically significant) will be summarised for each visit, by treatment group and overall.

#### 11.12. Endocrinology

The following will be summarised for each visit (as appropriate) by treatment group and overall.

- Female breast development and pubic hair development.
- Male testicular volume, genital development and pubic hair development.
- Change from baseline in male testicular volume.
- Change from baseline in plasma endocrine parameters (Follicle Stimulating Hormone, Luteinizing Hormone, Sex Hormone Binding Globulin, Total Testosterone and Inhibin B) by gender.

The above tables will also be summarised by pubertal status at baseline defined as follows:

Male: Pre-pubertal: testicular volume  $\leq 4$  ml, Post-pubertal: testicular volume  $\geq 4$  ml.

Female: Pre-pubertal: Stage 1 breast development, Post-pubertal: Stage  $\geq 2$  breast development.

## 11.13. Pregnancies (as applicable)

A listing of pregnancy events will be provided, as necessary.

#### 12. EFFICACY ANALYSES

Efficacy data will be presented for the Intent-to-Treat Population unless otherwise specified.

The following will be summarised for observed case data for each visit (as appropriate) by treatment group and overall.

- The absolute value, change from baseline and % change from baseline in the 6 minute walking distance (6MWD) test, overall and by oxygen use.
- The walking duration for subjects who walked less than six minutes.
- The use of oxygen during the 6MWD test.
- The time to clinical worsening of PAH.
- The criteria for clinical worsening of PAH.
- WHO Functional Class and change from baseline in WHO Functional Class.
- The absolute value and percent change from baseline, using log-transformed data, in N-terminal pro-B-type natriuretic peptide (NT-Pro BNP) concentration.
- The absolute value and change from baseline in the number of school days, missed school days and missed school days due to PAH.

 The absolute value and change from baseline in Subject Global Assessment as measured by the SF-10 health survey for children and summarised for the physical summary score (PHS-10) and the psychosocial summary score (PSS-10).

Further table will be produced summarizing change in WHO FC scores categorized in terms of "-2, -1, 0, +1, +2" and in terms of "Improved, No Change, Deteriorated" (see Section 9.2.3 and Section 9.2.4).

#### 12.1. Exploratory analyses

The following will be summarised for each visit, by treatment group and overall.

The absolute value and change from baseline in exploratory echocardiogram:pericardial effusion, right atrial pressure, tricuspid annular plane systolic excursion, eccentricity index (systolic and diastolic), tricuspid regurgitant jet velocity and right ventricular pressure.

#### 12.2. Other analyses

The following will be summarised for each visit, by treatment group and overall.

The absolute value and change from baseline in cardiopulmonary hemodynamics (at centres where the collection of hemodynamic data is considered part of the standard of care):- heart rate, mean arterial blood pressure, mean pulmonary arterial pressure, mean right atrial pressure, left ventricular end diastolic pressure or pulmonary capillary wedge pressure, pulmonary vascular resistance, cardiac output, cardiac index (calculated value), arterial oxygen saturation and mixed venous oxygen saturation.

#### 13. CLINICAL PHARMACOLOGY DATA ANALYSES

## 13.1. Pharmacokinetic Analyses

Not applicable.

## 13.2. Pharmacodynamic Analyses

Not applicable.

## 13.3. Pharmacokinetic/Pharmacodynamic Analyses

Not applicable.

#### 14. BIOMARKER DATA ANALYSIS

Not applicable.

#### 15. PHARMACOGENETIC DATA ANALYSES

Not applicable.

## 16. VIRAL GENOTYPING/PHENOTYPING

Not applicable.

## 17. REFERENCES

Not Applicable.

## 18. ATTACHMENTS

## 18.1. Table of Contents for Data Display Specifications

## 18.1.1. Tables

Table numbering for the Japanese subgroup will be add 001 at the end of the table number. Thus, Table 1.1 will become 1.1001. Table numbering for the Age Strata subgroup will be add 002 at the end of the table number. Thus, Table 1.5 will become 1.5002.

Population Tables

| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 1.1 | Summary of Subject Disposition | Intent-to-<br>Treat | 1.1 | X | | Interim, SAC |
| 1.2 | Summary of Study Populations | Randomised | 1.2 | | | Interim, SAC |
| 1.3 | Summary of Subjects by Country and Centre | Intent-to-<br>Treat | 1.3 | | | Interim, SAC |
| 1.4 | Summary of Inclusion/Exclusion Criteria Deviations | Intent-to-<br>Treat | 1.4 | | | Interim, SAC |
| 1.5 | Summary of Demographic and Baseline Characteristics | Intent-to-<br>Treat | 1.5 | X | Х | Interim, SAC |
| 1.6 | Summary of Past Medical Conditions | Intent-to-<br>Treat | 1.6 | | Х | Interim, SAC |
| 1.7 | Summary of Current Medical Conditions | Intent-to-<br>Treat | 1.6 | | Х | Interim, SAC |
| 1.8 | Summary of Concomitant Medications | Intent-to-<br>Treat | 1.8 | X | | Interim, SAC |
| 1.9 | Summary of Ongoing Background PAH Therapy at Baseline<br>By Drug Class and Preferred Term | Intent-to-<br>Treat | 1.9 | | X | Interim, SAC |
| 1.10 | Summary of Ongoing Background PAH Therapy at Week 24 By Drug Class and Preferred Term | Intent-to-<br>Treat | 1.9 | | Х | Interim, SAC |
| 1.11 | Summary of Subjects who continue in the long term study (AMB 114588) | Intent-to-<br>Treat | 1.11 | | | Interim, SAC |

#### AMB112529

| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 1.12 | Summary of Compliance to Investigational Product since last visit | Intent-to-<br>Treat | 1.12 | | | Interim, SAC |
| 1.13 | Summary of Investigational Product Compliance Overall | Intent-to-<br>Treat | 1.13 | | | Interim, SAC |
| 1.14 | Summary of Important Protocol Deviation | Intent-to-<br>Treat | 1.14 | | | Interim, SAC |

## Efficacy Tables

| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 2.1 | Summary of 6 Minute Walking Distance (meters) | Intent-to-<br>Treat | 2.1 | X | X | Interim, SAC |
| 2.2 | Summary of Change from Baseline in 6 Minute Walking Distance (meters) | Intent-to-<br>Treat | 2.1 | Х | X | Interim, SAC |
| 2.3 | Summary of Percent Change from Baseline in 6 Minute Walking Distance (meters) | Intent-to-<br>Treat | 2.1 | Х | X | Interim, SAC |
| 2.4 | Summary of Walking Duration (minutes) for subjects who walked less than six minutes | Intent-to-<br>Treat | 2.4 | Х | X | Interim, SAC |
| 2.5 | Summary of use of Oxygen during 6 Minute Walking exercise (L/min) | Intent-to-<br>Treat | 2.5 | Х | X | Interim, SAC |
| 2.6 | Summary of Time to Clinical Worsening of PAH (days) | Intent-to-<br>Treat | 2.6 | Х | | Interim, SAC |
| 2.7 | Summary of Clinical Worsening of PAH | Intent-to-<br>Treat | 2.7 | | | Interim, SAC |
| 2.8 | Summary of WHO Functional Class | Intent-to-<br>Treat | 2.8 | X | X | Interim, SAC |
| 2.9 | Summary of Change from Baseline in WHO Functional Class | Intent-to-<br>Treat | 2.8 | Х | Х | Interim, SAC |

| | | T | | 1 | 1 | AMB112529 |
|---|---|---|---|---|---|---|
| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
| 2.10 | Summary of WHO Functional Class Shifts from Baseline by Visit | Intent-to-<br>Treat | 2.10 | X | X | Interim, SAC |
| 2.11 | Summary of WHO Functional Class Change from Baseline Categorisation | Intent-to-<br>Treat | 2.11 | X | Х | Interim, SAC |
| 2.12 | Summary of Plasma NT-Pro BNP concentration (ng/L) | Intent-to-<br>Treat | 2.12 | Х | X | Interim, SAC |
| 2.13 | Summary of Ratio to Baseline in Plasma NT-Pro BNP concentration (%) | Intent-to-<br>Treat | 2.12 | X | X | Interim, SAC |
| 2.14 | Summary of Exploratory Echocardiogram | Intent-to-<br>Treat | 2.14 | X | X | Interim, SAC |
| 2.15 | Summary of Change from Baseline in Exploratory Echocardiogram | Intent-to-<br>Treat | 2.15 | X | X | Interim, SAC |
| 2.16 | Summary of Cardiopulmonary Hemodynamics | Intent-to-<br>Treat | 2.16 | Х | | Interim, SAC |
| 2.17 | Summary of Change from Baseline in Cardiopulmonary Hemodynamics | Intent-to-<br>Treat | 2.16 | Х | | Interim, SAC |
| 2.18 | Summary of Number of Subjects with School Days within the Past Month | Intent-to-<br>Treat | 2.18 | X | X | Interim, SAC |
| 2.19 | Summary Statistics of School Days within the past month | Intent-to-<br>Treat | 2.19 | X | X | Interim, SAC |
| 2.20 | Summary Statistics of Change from Baseline in School Days within the Past month | Intent-to-<br>Treat | 2.19 | X | X | Interim, SAC |
| 2.21 | Summary of Subject Global Assessment (SF10 Health Survey for Children) | Intent-to-<br>Treat | 2.21 | X | X | Interim, SAC |
| 2.22 | Summary of Change from Baseline in Subject Global Assessment (SF10 Health Survey for Children) | Intent-to-<br>Treat | 2.21 | X | X | Interim, SAC |
| 2.23 | Summary of SF10 Health Survey - Number and Percentage of Subjects with Particular Item Responses | Intent-to-<br>Treat | 2.23 | X | X | Interim, SAC |

#### Safety Tables

| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 3.1 | Summary of Exposure to Investigational Product | Safety | 3.1 | X | X | Interim, SAC |
| 3.2 | Summary of Treatment-Emergent Adverse Events | Safety | 3.2 | Х | Х | Interim, SAC |
| 3.3 | Summary of Treatment-Emergent Adverse Events by Preferred Term | Safety | 3.3 | | X | Interim, SAC |
| 3.4 | Summary of Treatment-Emergent Adverse Events by Maximum Intensity | Safety | 3.4 | Х | | Interim, SAC |
| 3.5 | Summary of Treatment-Emergent Adverse Events by Action Taken with IP | Safety | 3.5 | | | Interim, SAC |
| 3.6 | Summary of Treatment-Emergent Adverse Events leading to Permanent Discontinuation of IP or Withdrawal from the Study | Safety | 3.2 | | X | Interim, SAC |
| 3.7 | Summary of Treatment-Emergent Adverse Events related to IP | Safety | 3.2 | Х | Х | Interim, SAC |
| 3.8 | Summary of Cumulative Incidence of Treatment-Emergent Adverse Events by Time to First Occurrence | Safety | 3.8 | | | Interim, SAC |
| 3.9 | Summary of Serious Treatment-Emergent Adverse Events | Safety | 3.2 | | Х | Interim, SAC |
| 3.10 | Summary of Serious Treatment-Emergent Adverse Events - Number of Subjects and Occurrences | Safety | 3.10 | | | Interim, SAC |
| 3.11 | Summary of Serious Treatment-Emergent Adverse Events by Outcome | Safety | 3.11 | | | Interim, SAC |
| 3.12 | Summary of Serious Treatment-Emergent Adverse Events by Action Taken with IP | Safety | 3.5 | | | Interim, SAC |
| 3.13 | Summary of Serious Treatment-Emergent Adverse Events leading to Permanent Discontinuation of IP or Withdrawal from the Study | Safety | 3.2 | | | Interim, SAC |
| 3.14 | Summary of Serious Treatment-Emergent Adverse Events related to IP | Safety | 3.2 | | | Interim, SAC |
| 3.15 | Summary of Fatal Serious Treatment-Emergent Adverse Events | Safety | 3.2 | | | Interim, SAC |
| 3.16 | Summary of Fatal Serious Treatment-Emergent Adverse Events related to IP | Safety | 3.2 | | | Interim, SAC |

| | T | | | | | AMB112529 |
|---|---|---|---|---|---|---|
| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
| 3.17 | Summary of Treatment-Emergent Adverse Events of Special Interest | Safety | 3.2 | X | | Interim, SAC |
| 3.18 | Summary of Treatment-Emergent Adverse Events of Special Interest leading to Permanent Discontinuation of IP or Withdrawal from the Study | Safety | 3.2 | | | Interim, SAC |
| 3.19 | Summary of Cumulative Incidence of Treatment-Emergent<br>Adverse Events of Special Interest by Time to First<br>Occurrence | Safety | 3.8 | | | Interim, SAC |
| 3.20 | Summary of Most Common (>5%) Non-Serious Treatment-<br>Emergent Adverse Events - Number of Subjects and<br>Occurrences | Safety | 3.10 | | | Interim, SAC |
| 3.21 | Summary of Haematology Data | Safety | 3.21 | Х | | Interim, SAC |
| 3.22 | Summary of Change from Baseline in Haematology Data | Safety | 3.21 | Х | | Interim, SAC |
| 3.23 | Summary of Haematology Data of Potential Clinical Concern | Safety | 3.23 | X | | Interim, SAC |
| 3.24 | Summary of Clinical Chemistry Data | Safety | 3.21 | Х | | Interim, SAC |
| 3.25 | Summary of Change from Baseline in Clinical Chemistry Data | Safety | 3.21 | X | | Interim, SAC |
| 3.26 | Summary of Clinical Chemistry Data of Potential Clinical Concern | Safety | 3.23 | Х | | Interim, SAC |
| 3.27 | Summary of Endocrinology Laboratory Data (females only) | Safety | 3.21 | Х | | Interim, SAC |
| 3.28 | Summary of Change from Baseline in Endocrinology Laboratory Data (females only) | Safety | 3.21 | Х | | Interim, SAC |
| 3.29 | Summary of Liver Events Assessment | Safety | 3.29 | | | Interim, SAC |
| 3.30 | Summary of Vital Signs | Safety | 3.30 | X | | Interim, SAC |
| 3.31 | Summary of Change from Baseline in Vital Signs | Safety | 3.30 | X | | Interim, SAC |
| 3.32 | Summary of Vital Signs Data of Potential Clinical Concern | Safety | 3.32 | X | | Interim, SAC |

| m 1 1 | m1. 3 | I | I | T - | | |
|---|---|---|---|---|---|---|
| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
| 3.33 | Summary of Change from Baseline in Vital Signs Data of Potential Clinical Concern | Safety | 3.32 | X | | Interim, SAC |
| 3.34 | Summary of Physical Examination by Visit | Safety | 3.34 | Х | | Interim, SAC |
| 3.35 | Summary of 12-lead ECG | Safety | 3.35 | Х | | Interim, SAC |
| 3.36 | Summary of Endocrinology assessments by Visit - Female | Safety | 3.36 | X | | Interim, SAC |
| 3.37 | Summary of Endocrinology assessments by Visit - Male | Safety | 3.37 | Х | | Interim, SAC |
| 3.38 | Summary of Pubertal Development Shifts from Baseline - Female | Safety | 3.38 | X | | Interim, SAC |
| 3.39 | Summary of Pubertal Development Shifts from Baseline - Male | Safety | 3.39 | X | | Interim, SAC |
| 3.40 | Summary of Testicular Volume Change from Baseline - Male | Safety | 3.40 | X | | Interim, SAC |
| 3.41 | Summary of Change from Baseline in Plasma Endocrine<br>Parameters - Female | Safety | 3.41 | X | | Interim, SAC |
| 3.42 | Summary of Change from Baseline in Plasma Endocrine<br>Parameters - Male | Safety | 3.42 | X | | Interim, SAC |

## **18.1.2.** Listings

Population Listings

| Listing<br>Number | Title | Population | Template<br>Listing | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 1.1 | Listing of Randomised and Actual Treatments | Intent-to-<br>Treat | 1.1 | | | Interim, SAC |
| 1.2 | Listing of Reasons for Study Withdrawal | Intent-to-<br>Treat | 1.2 | | | Interim, SAC |
| 1.3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | Intent-to-<br>Treat | 1.3 | | | Interim, SAC |
| 1.4 | Listing of Demographic Characteristics | Intent-to-<br>Treat | 1.4 | | | Interim, SAC |
| 1.5 | Listing of Race | Intent-to-<br>Treat | 1.5 | | | Interim, SAC |
| 1.6 | Listing of Disease History | Intent-to-<br>Treat | 1.6 | | | Interim, SAC |
| 1.7 | Listing of Medical Conditions | Intent-to-<br>Treat | 1.7 | | | Interim, SAC |
| 1.8 | Listing of Medications | Intent-to-<br>Treat | 1.8 | | | Interim, SAC |
| 1.9 | Listing of PAH Therapy | Intent-to-<br>Treat | 1.9 | | | Interim, SAC |
| 1.10 | Relationship between ATC Level 1, Ingredient and Verbatim Text | Intent-to-<br>Treat | 1.10 | | | Interim, SAC |
| 1.11 | Listing of Protocol Deviation | Intent-to-<br>Treat | 1.11 | | | Interim, SAC |

## Efficacy Listings

| Listing<br>Number | Title | Population | Template<br>Listing | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup | Deliverable |
|---|---|---|---|---|---|---|
| 2.1 | Listing of 6 Minute Walk Distance Data | Intent-to-<br>Treat | 2.1 | | analysis | Interim, SAC |
| 2.2 | Listing of Clinical Worsening of PAH | Intent-to-<br>Treat | 2.2 | | | Interim, SAC |
| 2.3 | Listing of WHO Functional Class Data | Intent-to-<br>Treat | 2.3 | | | Interim, SAC |
| 2.4 | Listing of Plasma NT-Pro BNP Concentration (ng/L) | Intent-to-<br>Treat | 2.4 | | | Interim, SAC |
| 2.5 | Listing of Exploratory Echocardiogram | Intent-to-<br>Treat | 2.5 | | | Interim, SAC |
| 2.6 | Listing of Cardiopulmonary Hemodynamics | Intent-to-<br>Treat | 2.6 | | | Interim, SAC |
| 2.7 | Listing of School Days | Intent-to-<br>Treat | 2.7 | | | Interim, SAC |
| 2.8 | Listing of Subject Global Assessment (SF10 Health Survey for Children) | Intent-to-<br>Treat | 2.8 | | | Interim, SAC |

## Safety Listings

| Listing<br>Number | Title | Population | Template<br>Listing | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 3.1 | Listing of Exposure and Compliance to Investigational Product | Safety | 3.1 | | | Interim, SAC |
| 3.2 | Listing of All Adverse Events | Safety | 3.2 | | | Interim, SAC |
| 3.3 | Listing of Relationship between Adverse Event System Organ Class, Preferred Term and Verbatim Text | Safety | 3.3 | | | Interim, SAC |
| 3.4 | Listing of Subject Numbers for Specified Adverse<br>Events | Safety | 3.4 | | | Interim, SAC |
| 3.5 | Listing of Serious Adverse Events | Safety | 3.2 | | | Interim, SAC |

| Listing | Title | Population | Template | Japanese | Age | Deliverable |
|---|---|---|---|---|---|---|
| Number | | | Listing | subgroup<br>analysis | strata<br>subgroup<br>analysis | |
| 3.6 | Listing of Fatal Serious Adverse Events | Safety | 3.2 | | | Interim, SAC |
| 3.7 | Listing of Adverse Events Leading to Permanent<br>Discontinuation of Study Treatment or Withdrawal from<br>Study | Safety | 3.2 | | | Interim, SAC |
| 3.8 | Listing of Haematology | Safety | 3.8 | | | Interim, SAC |
| 3.9 | Listing of Haematology Data for Subjects with<br>Abnormalities of Potential Clinical Concern | Safety | 3.9 | | | Interim, SAC |
| 3.10 | Listing of Clinical Chemistry | Safety | 3.8 | | | Interim, SAC |
| 3.11 | Listing of Clinical Chemistry Data for Subjects with Abnormalities of Potential Clinical Concern | Safety | 3.9 | | | Interim, SAC |
| 3.12 | Listing of Endocrinology Laboratory Data - Females only | Safety | 3.8 | | | Interim, SAC |
| 3.13 | Listing of Liver Event Results and Time of Event Relative to Treatment | Safety | 3.13 | | | Interim, SAC |
| 3.14 | Listing of patient specific information for liver events | Safety | 3.14 | | | Interim, SAC |
| 3.15 | Listing of Medical Conditions for Subjects with Liver Events on Treatment | Safety | 3.15 | | | Interim, SAC |
| 3.16 | Listing of Liver Biopsy Details | Safety | 3.16 | | | Interim, SAC |
| 3.17 | Listing of Liver Imaging Details | Safety | 3.17 | | | Interim, SAC |
| 3.18 | Listing of Vital Signs | Safety | 3.18 | | | Interim, SAC |
| 3.19 | Listing of Vital Signs Data for Subjects with<br>Abnormalities of Potential Clinical Concern | Safety | 3.9 | | | Interim, SAC |
| 3.20 | Listing of Physical Examination | Safety | 3.20 | | | Interim, SAC |
| 3.21 | Listing of 12-Lead ECG Findings | Safety | 3.21 | | | Interim, SAC |
| 3.22 | Listing of Endocrinology Assessments | Safety | 3.22 | | | Interim, SAC |

| Listing | Title | Population | Template | Japanese | Age | Deliverable |
|---|---|---|---|---|---|---|
| Number | | | Listing | subgroup<br>analysis | strata<br>subgroup | |
| | | | | <del>-</del> | analysis | |
| 3.23 | Listing of Pregnancy Results | Safety | 3.23 | | | Interim, SAC |

## 18.1.3. Figures

Population Figures

| Figure<br>Number | Title | Population | Template<br>Figure | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 1.1 | Summary of Subject Accrual | Intent-to-<br>Treat | 1.1 | | _ | Interim, SAC |

## Efficacy Figures

| Figure<br>Number | Title | Population | Template<br>Figure | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 2.1 | Box plots of 6 Minute Walking Distance (meters) by Week | Intent-to-<br>Treat | 3.4 | | | Interim, SAC |
| 2.2 | Box plots of Change from Baseline in 6 Minute Walking Distance (meters) by Week | Intent-to-<br>Treat | 3.4 | | | Interim, SAC |
| 2.3 | Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to First Clinical Worsening of PAH | Intent-to-<br>Treat | 3.1 | | | Interim, SAC |
| 2.6 | Box plots of Plasma NT-Pro BNP concentration by Week | Intent-to-<br>Treat | 3.4 | | | Interim, SAC |
| 2.7 | Box plots of Change from Baseline in Plasma NT-Pro BNP concentration by Week | Intent-to-<br>Treat | 3.4 | | | Interim, SAC |
| 2.8 | Box plots of Exploratory Echocardiogram Data by Week | Intent-to-<br>Treat | 3.4 | X (Line plots of Explorato ry Echocardi ogram Data by Subject) see | | Interim, SAC |

| Figure<br>Number | Title | Population | Template<br>Figure | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| | | | | template 3.11) | | |
| 2.9 | Box plots of Change from Baseline in Exploratory<br>Echocardiogram Data by Week | Intent-to-<br>Treat | 3.5 | | | Interim, SAC |

## Safety Figures

| Figure<br>Number | Title | Population | Template<br>Figure | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 3.1 | Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to First Treatment-Emergent Adverse Event | Safety | 3.1 | | - | Interim, SAC |
| 3.2 | Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to First Serious Adverse Event | Safety | 3.1 | | | Interim, SAC |
| 3.3 | Bar Chart of Treatment-Emergent Adverse Events Occurring in Two or More Subjects in any Treatment Group | Safety | 3.3 | | | Interim, SAC |
| 3.4 | Box plots of Haematology Data by Week (Selected Parameters) | Safety | 3.4 | | | Interim, SAC |
| 3.5 | Box plots of Change from Baseline in Haematology Data by Week (Selected Parameters) | Safety | 3.4 | | | Interim, SAC |
| 3.6 | Box plots of Chemistry Data by Week (Selected Parameters) | Safety | 3.4 | | | Interim, SAC |
| 3.7 | Box plots of Change from Baseline in Chemistry Data by Week (Selected Parameters) | Safety | 3.4 | | | Interim, SAC |
| 3.8 | Patient Profiles of Liver Function Tests | Safety | 3.8 | | | Interim, SAC |
# CONFIDENTIAL

## AMB112529

| Figure<br>Number | Title | Population | Template<br>Figure | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 3.9 | Box plots of Vital Signs Data by Week | Safety | 3.4 | | | Interim, SAC |
| 3.10 | Box plots of Change from Baseline in Vital Signs Data by Week | Safety | 3.4 | | | Interim, SAC |
| 3.11 | Line plots of Endocrinology Assessments by subject | Safety | 3.11 | | | Interim, SAC |

# 18.2. Data Display Specifications

Protocol: AMB112529 Page 1 of n

Population: Intent-to-Treat

Table 1.1: Summary of Subject Disposition

| | Ambrise<br>Low Dos<br>(N=XXX) | | Ambrise<br>High Do<br>(N=XXX) | ose | Total<br>(N=XXX) | |
|---|---|---|---|---|---|---|
| Subject status | | | | | | |
| Completed | XX | (%) | XX | (%) | XX | (%) |
| Withdrawn | XX | (%) | XX | (%) | XX | (%) |
| Died | | | | | | |
| Primary reason for study withdrawal * | | | | | | |
| Adverse event | XX | (%) | XX | (%) | XX | (%) |
| Lack of Efficacy | XX | (%) | XX | (%) | XX | (%) |
| Protocol Deviation | XX | (%) | XX | (%) | XX | (%) |
| Subject reached protocol defined stopping criteria | XX | (%) | XX | (%) | XX | (응) |
| Study closed/terminated | XX | (%) | XX | (%) | XX | (%) |
| Lost to Follow-up | XX | (%) | XX | (%) | XX | (%) |
| Investigator discretion | XX | (%) | XX | (%) | XX | (%) |
| Withdrew consent | XX | (%) | XX | (%) | XX | (%) |

Note: \* Percentages are based on the number of subjects in the treatment group. Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Programming notes: Denominator for each primary reason for withdrawal is number of subjects in the Intent-to-Treat population per treatment group.

Protocol: AMB112529
Population: Randomised

Table 1.2: Summary of Study Populations

| | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Randomised | XXX | XXX | XXX |
| Safety Population | XXX (%) | XXX (%) | XXX (%) |
| Intention-to-Treat population | XXX (%) | XXX (%) | XXX (%) |

Note: The Safety Population is defined as all randomized subjects who received at least 1 dose of study drug. Subjects are considered as belonging to the treatment group according to highest dose received. The Intention-to-Treat (ITT) Population is defined as all randomized subjects who received at least 1 dose of study drug. Subjects are considered as belonging to their randomized treatment group, regardless of the actual dose of ambrisentan received.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: See notes above relating to denominators for percentages.

Population: Intent-to-treat

Table 1.3: Summary of Subjects by Country and Centre

| Country | Centre ID | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|
| XXXXXXXX | All<br>XXXXXX | XX (%)<br>XX (%) | XX (%)<br>XX (%) | XX (%)<br>XX (%) |
| XXXXXXXX | All | XX (%) | XX (%) | XX (%) |
| | XXXXXX | XX (%) | XX (%) | XX (%) |
| XXXXXXXX | All | XX (%) | XX (%) | XX (%) |
| | XXXXXX | XX (%) | XX (%) | XX (%) |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Population: Intent-to-Treat

Table 1.4: Summary of Inclusion/Exclusion Criteria Deviations

| | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Any criteria deviations | XX (%) | XX (%) | XX (%) |
| Inclusion I1 I2 Etc | XX (%)<br>XX (%) | XX (%)<br>XX (%) | XX (%)<br>XX (%) |
| Exclusion E1 E2 Etc | XX (%)<br>XX (%) | XX (%) | XX (%)<br>XX (%) |

Note: Please refer to numbering of inclusion and exclusion criteria in protocol. Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Programming notes: Only present criteria where there is at least one (total) deviation. "Any criteria deviations" is the number of subjects who had at least one deviation.

Population: Intent-to-Treat

Table 1.5: Summary of Demographic and Baseline Characteristics

| | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Age (yrs) | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |
| Age (yrs) | | | |
| n | XXX | XXX | XX (%) |
| <8 years | XX (%) | XX (%) | XX (%) |
| 8 - 11 years | XX (%) | XX (%) | XX (%) |
| 12 - <18 years | XX (%) | XX (%) | XX (%) |
| >=18 years | XX (%) | XX (%) | XX (%) |
| Sex | | | |
| n | XXX | XXX | XX (%) |
| Female | XX (%) | XX (%) | XX (%) |
| Male | XX (%) | XX (%) | XX (%) |

Note: \* A subject may be represented in more than one geographic ancestry group. Q1 = 1st quartile, Q3 = 3rd quartile. Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

CONFIDEN

Protocol: AMB112529

Population: Intent-to-Treat

Table 1.5: Summary of Demographic and Baseline Characteristics

| | Ambrisent<br>Low Dose<br>(N=XXX) | tan | Ambrisent<br>High Dose<br>(N=XXX) | - | Total<br>(N=XXX) | |
|---|---|---|---|---|---|---|
| Child Bearing Potential (Females only) | | | | | | |
| n | XXX | | XXX | | XXX | |
| Pre-menarcheal | XX | (응) | XX | (%) | XX | (응) |
| Sterile (of child bearing age) | XX | (%) | XX | (%) | XX | (%) |
| Potentially able to bear children | XX | (응) | XX | (%) | XX | (응) |
| Ethnicity | | | | | | |
| n | XXX | | XXX | | XXX | |
| Hispanic/Latino | XX | (응) | XX | (%) | XX | (%) |
| Not Hispanic/Latino | XX | (%) | XX | (%) | XX | (%) |
| Geographic Ancestry | | | | | | |
| n | XXX | | XXX | | XXX | |
| African American/African Heritage | XX | (%) | XX | (응) | XX | (응) |
| American Indian or Alaskan Native | XX | (응) | XX | (응) | XX | (응) |
| Asian - Central/South Asian Heritage | XX | (%) | XX | (응) | XX | (응) |
| Asian - East Asian Heritage | XX | (%) | XX | (응) | XX | (응) |
| Asian - Japanese Heritage | XX | (응) | XX | (응) | XX | (응) |
| Asian - South East Asian Heritage | XX | (응) | XX | (응) | XX | (응) |
| Native Hawaiian or Other Pacific Islander | XX | (%) | XX | (%) | XX | (%) |
| White - Arabic/North African Heritage | XX | (%) | XX | (%) | XX | (응) |
| White - White/Caucasian/European Heritage | XX | (%) | XX | (%) | XX | (%) |

Note: \* A subject may be represented in more than one geographic ancestry group. Q1 = 1st quartile, Q3 = 3rd quartile. Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

CONTIDE

Population: Intent-to-Treat

Protocol: AMB112529

Table 1.5: Summary of Demographic and Baseline Characteristics

| | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Weight (kg) | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |
| Weight (kg) | | | |
| n | XXX | XXX | XX (%) |
| <20 kg | XX (%) | XX (%) | XX (%) |
| 20 - <35 kg | XX (%) | XX (%) | XX (%) |
| 35 <b>-</b> <50 kg | XX (%) | XX (%) | XX (%) |
| >=50 kg | XX (%) | XX (%) | XX (%) |
| Aetiology of PAH Randomised Strata | | | |
| n | XXX | XXX | XX (%) |
| Idiopathic (IPAH) | XX (%) | XX (%) | XX (%) |
| Familial (FPAH) | XX (%) | XX (%) | XX (%) |
| Persistent PAH despite surgical repair | XX (%) | XX (%) | XX (%) |
| Secondary to connective tissue disease | XX (%) | XX (%) | XX (%) |

Note: \* A subject may be represented in more than one geographic ancestry group.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Population: Intent-to-Treat

Table 1.5: Summary of Demographic and Baseline Characteristics

| | Ambrisentan<br>Low Dose | Ambrisentan<br>High Dose | Total<br>(N=XXX) |
|---|---|---|---|
| | (N=XXX) | (N=XXX) | |
| Duration of PAH (days) | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |
| PAH Therapy Use | | | |
| n | XXX | XXX | XX (%) |
| Ongoing PAH therapy at baseline | XX (%) | XX (%) | XX (%) |
| Prior PAH therapy, not ongoing at baseline | XX (%) | XX (%) | XX (%) |
| No PAH therapy recorded | XX (%) | XX (%) | XX (%) |

Note: \* A subject may be represented in more than one geographic ancestry group.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Population: Intent-to-Treat

Table 1.5: Summary of Demographic and Baseline Characteristics

| | 7.1.1 | 7 1 1 | m |
|------------------------|-------------|-------------|---------|
| | Ambrisentan | Ambrisentan | Total |
| | Low Dose | High Dose | (N=XXX) |
| | (N=XXX) | (N=XXX) | |
| NUO Eurobianal Class | | | |
| WHO Functional Class | | | |
| N | XXX | XXX | XX (%) |
| Class II | XX (%) | XX (%) | XX (%) |
| Class III | XX (%) | XX (%) | XX (%) |
| 6 minute walk data (m) | | | |
| N | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |

Note: \* A subject may be represented in more than one geographic ancestry group.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

CONTIDE

Population: Intent-to-Treat

Protocol: AMB112529

Table 1.6: Summary of Past Medical Conditions

| Classification | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Any condition | XX (%) | XX (%) | XX (%) |
| Classification 1 Any condition Preferred Term 1 Preferred Term 2 etc | XX (%) | XX (%) | XX (%) |
| | XX (%) | XX (%) | XX (%) |
| | XX (%) | XX (%) | XX (%) |
| Classification 2 Any condition Preferred Term 1 Preferred Term 2 etc | XX (%) | XX (%) | XX (%) |
| | XX (%) | XX (%) | XX (%) |
| | XX (%) | XX (%) | XX (%) |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Programming notes: "Any condition" relates to the number and percentage of subjects who had at least one condition. Subjects may be counted more than once across classifications.

Population: Intent-to-Treat

Protocol: AMB112529

Table 1.8: Summary of Concomitant Medications

| ATC Level 1 Preferred Term | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Any medication | XX (%) | XX (%) | XX (%) |
| Endocrine & Metabolic | | | |
| Any medication | XX (%) | XX (%) | XX (%) |
| Fluticasone propionate | XX (%) | XX (%) | XX (%) |
| Beclomethasone dipropionate | XX (%) | XX (%) | XX (%) |
| Anti-infectives & immunologicals | | | |
| Any medication | XX (%) | XX (%) | XX (%) |
| Amoxycillin | XX (%) | XX (%) | XX (%) |
| Amoxycillin trihydrate | XX (%) | XX (%) | XX (%) |
| Clamoxyl | XX (%) | XX (%) | XX (%) |
| Cefaclor | XX (%) | XX (%) | XX (%) |
| Cefproxil | XX (%) | XX (%) | XX (%) |

Etc..

Note: A medication may be included in more than one ATC level category and appear more than once. Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Programming notes: Medications will be sorted in descending order of total incidence across treatment groups for the ATC level 1 and in descending order of total incidence for the preferred term within each ATC level. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Population: Intent-to-Treat

Protocol: AMB112529

Table 1.9: Summary of Ongoing Background PAH Therapy at Baseline
By Drug Class and Preferred Term

| | Ambrisentan<br>Low Dose | Ambrisentan<br>High Dose | Total |
|---|---|---|---|
| PAH Therapy | (N=XXX) | (N=XXX) | (N=XXX) |
| Any medication | XX (%) | XX (%) | XX (%) |
| PDE5i (monotherapy) | | | |
| Any medication | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 | XX (%) | XX (%) | XX (%) |
| Etc | | | |
| Prostanoid (monotherapy) | | | |
| Any medication | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 | XX (%) | XX (%) | XX (%) |
| Etc | | | |
| PDE5i and prostanoid in combination | | | |
| Any medication | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 + Preferred Term 2 | XX (%) | XX (%) | XX (%) |
| Preferred Term 3 + Preferred Term 4 | XX (%) | XX (%) | XX (%) |
| Etc | | | |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Protocol: AMB112529
Population: Intent-to-Treat

Table 1.11: Summary of Subjects who continue in the long term study (AMB114588)

| Ambrisentan<br>Low Dose | Ambrisentan<br>High Dose | Total |
|---|---|---|
| (N=XXX) | (N=XXX) | (N=XXX) |
| XX (%) | XX (%) | XX (%)<br>XX (%) |
| | Low Dose<br>(N=XXX) | Low Dose High Dose (N=XXX) (N=XXX) |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Population: Intent-to-Treat

Table 1.12: Summary of Compliance to Investigational Product since last visit

| Planned Relative Time | Compliance assessment | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total |
|---|---|---|---|---|
| Flammed Relative lime | Compilance assessment | (IN-VVV) | (IN-VVV) | (IN-VVV) |
| Week 2 | n | XXX | XXX | XXX |
| | 0% compliant | XX (%) | XX (%) | XX (%) |
| | >0% and < 80% | XX (%) | XX (%) | XX (%) |
| | >= 80% and <= 120% | XX (%) | XX (%) | XX (%) |
| | >120% compliant | XX (%) | XX (%) | XX (%) |
| Week 4 | n | XXX | XXX | XXX |
| | 0% compliant | XX (%) | XX (%) | XX (%) |
| | >0% and < 80% | XX (%) | XX (%) | XX (%) |
| | >= 80% and <= 120% | XX (%) | XX (%) | XX (%) |
| | >120% compliant | XX (%) | XX (%) | XX (%) |
| Etc | Etc | | | |

Note: EW = Early Withdrawal.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>=35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Present for Weeks 2, 4, 8, 12, 16, 20, 24 and EW.

Population: Intent-to-treat

Table 1.13: Summary of Investigational Product Compliance Overall

| | Ambrisentan<br>Lose Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Overall % of visits at which subject is compliant | XX | XX | XX |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |

Note: Q1 = 1<sup>st</sup> quartile, Q3 = 3<sup>rd</sup> quartile.

Compliant visits are those at which subjects are  $\geq 80\%$  and  $\leq 120\%$  compliant. Compliance is determined by the site.

At a subject level compliance = 100\* (the number of visits at which the subject was compliant)/(the sum of all study visits for the subject). At a treatment group level the overall compliance = 100\* (the total number of visits at which all subjects in that group were compliant)/(the sum of all study visits for all subjects in that group).

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight >= 20 kg and <35 kg); 7.5 mg (>= 35 kg and <50 kg); 10 mg (>= 50 kg).

Protocol: AMB112529
Population: Intent-to-Treat

Table 1.14: Summary of Important Protocol Deviation

| | Ambrisentan<br>Low Dose | Ambrisentan<br>High Dose | Total |
|---|---|---|---|
| Protocol Deviation Category | (N=XXX) | (N=XXX) | (N=XXX) |
| Any Deviation | XX (%) | XX (%) | XX (%) |
| Eligibility criteria not met | XX (%) | XX (%) | XX (%) |
| Not withdrawn after developing withdrawal criteria | XX (%) | XX (%) | XX (%) |
| Prohibited medication or device | XX (%) | XX (%) | XX (%) |
| Visit window | XX (%) | XX (%) | XX (%) |
| Informed consent procedure | XX (%) | XX (%) | XX (%) |
| Administer/dispense study medication | XX (%) | XX (%) | XX (%) |
| Failure to report SAE, Pregnancy, or liver function abnormalities per protocol | XX (%) | XX (%) | XX (%) |
| Study blind/ unblind procedures | XX (%) | XX (%) | XX (%) |
| Study treatment supply procedures | XX (%) | XX (%) | XX (%) |
| Biological specimen sample procedures | XX (%) | XX (%) | XX (%) |
| Assessment procedures | XX (%) | XX (%) | XX (%) |
| Diary Card procedures | XX (%) | XX (%) | XX (%) |
| Equipment procedures | XX (%) | XX (%) | XX (%) |
| Randomization procedures | XX (%) | XX (%) | XX (%) |
| Other | XX (%) | XX (%) | XX (%) |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

33.11.12

Population: Intent-to-Treat

Protocol: AMB112529

Table 2.1: Summary of 6 Minute Walking Distance (meters)

| Treatment | Planned | n | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| | Relative Time | | | | | | | | |
| Ambrisentan | Baseline* | | | | | | | | |
| Low Dose | Overall | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | With oxygen use | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Without oxygen use | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | Week 4 | | | | | | | | |
| | Overall | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | With oxygen use | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Without oxygen use | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Etc | | | | | | | | |
| | Week 24 | | | | | | | | |
| | EW | | | | | | | | |
| Ambrisentan | Etc | | | | | | | | |
| High Dose | | | | | | | | | |
| (N=XXX) | | | | | | | | | |
| Total | Etc | | | | | | | | |
| (N=XXX) | | | | | | | | | |
| , | | | | | | | | | |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>=35 kg).

High dose, 5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ =35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ =50 kg).

Population: Intent-to-Treat

Table 2.4: Summary of Walking Duration (minutes) for subjects who walked less than six minutes

| Treatment | Number of subjects who attempted the 6 minute walk | Planned<br>Relative Time | n | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| Ambrisentan | | Baseline* | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Low Dose | | | | | | | | | | |
| (N=XXX) | | Week 4 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 8 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 12 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 16 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 20 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 24 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | EW | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Ambrisentan<br>High Dose | | Baseline* | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | | Week 4 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 8 | XX (%) | | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 12 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 16 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 20 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 24 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | EW | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Total | | Etc | | | | | | | | |

(N=XXX)

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

% out of the number of subjects who attempted the 6 minute walk.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

Population: Intent-to-Treat

Table 2.5: Summary of use of Oxygen during 6 Minute Walking exercise (L/min)

| Treatment | Number of subjects who attempted the 6 minute walk | Planned<br>Relative Time | n | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| Ambrisentan<br>Low Dose | | Baseline* | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | | Week 4 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (IN-VVV) | | Week 4<br>Week 8 | XX (%)<br>XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | | ` , | | XX.XX | | | XX.X | XX | |
| | | Week 12 | XX (%) | XX.X | | XX.X | XX.X | | XX | XX |
| | | Week 16 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | | XX |
| | | Week 20 | XX (%) | XX.X | XX.XX | XX.X | XX . X | XX.X | XX | XX |
| | | Week 24 | XX (%) | XX.X | XX.XX | XX.X | XX . X | XX.X | XX | XX |
| | | EW | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Ambrisentan<br>High Dose | | Baseline* | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | | Week 4 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| , | | Week 8 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 12 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 16 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 20 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 24 | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | EW | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Total<br>(N=XXX) | Etc | | | | | | | | |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion. % out of the number of subjects who attempted the 6 minute walk.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

Population: Intent-to-Treat

Table 2.6: Summary of Time to the first Clinical Worsening of PAH (days)

| | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| N | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |

Note: Q1 = 1st quartile, Q3 = 3rd quartile. Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Table 2.7: Summary of Clinical Worsening of PAH

| | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Subjects with at least one criteria | XX (%) | XX (%) | XX (%) |
| Death (all cause) or placed on active list for lung transplant | XX (%) | XX (%) | XX (%) |
| Hospitalisation for worsening of PAH | XX (%) | XX (%) | XX (%) |
| Addition/increased dose of other targeted PAH therapetic agents and/or atrial septostomy | XX (%) | XX (%) | XX (%) |
| PAH related deterioration | XX (%) | XX (%) | XX (%) |
| PAH related deterioration:- | | | |
| Increase from baseline in WHO functional class | XX (%) | XX (%) | XX (%) |
| Deterioration in exercise testing | XX (%) | XX (%) | XX (%) |
| Clinical signs or symptoms of right sided heart failure | XX (%) | XX (%) | XX (%) |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Population: Intent-to-Treat

Population: Intent-to-Treat

Table 2.8: Summary of WHO Functional Class

| Treatment | Planned<br>Relative Time | n | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Ambrisentan<br>Low Dose | Baseline* | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | Week 4 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 8 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 12 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 16 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 20 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 24 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | EW | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Ambrisentan<br>High Dose | Baseline* | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | Week 4 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 8 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 12 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 16 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 20 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 24 | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | EW | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Total (N=XXX) | Etc | | | | | | | | |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There are 4 grades of WHO FC based on symptom severity (Class I=none, Class IV=most severe).

Grades mapped to numeric scale 1-4 (i.e. Class IV=4).

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion. EW = Early Withdrawal.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

#### PPD

Programming notes: Present Baseline and Weeks 4, 8, 12, 16, 20, 24 and EW.

Population: Intent-to-Treat

Table 2.10: Summary of WHO Functional Class Shifts from Baseline by Visit

| Treatment | Planned<br>Relative<br>Time | WHO<br>Functional<br>Class | Functional WHO Functional C | |
|---|---|---|---|---|
| | | _ | II | III |
| Ambrisentan Low Dose (N=XXX) | Week 4 | I | XX (%) | XX (%) |
| | | II<br>III | XX (%)<br>XX (%) | XX (%)<br>XX (%) |
| | | IV | XX (%) | XX (%) |
| | | Unknown/<br>Not Recorded | XX | XX |
| | Week 8 | I | XX (%) | XX (%) |
| | | II | XX (%) | XX (%) |
| | | III | XX (%) | XX (%) |
| | | IV | XX (%) | XX (%) |
| | | Unknown/<br>Not Recorded | XX | XX |

Etc..

Note: Baseline is the last value recorded prior to start of study treatment.

There are 4 grades of WHO FC based on symptom severity (Class I=none, Class IV=most severe).

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Present Weeks 4, 8, 12, 16, 20, 24 and EW, for each treatment group and overall.

Population: Intent-to-Treat

Protocol: AMB112529

Table 2.11: Summary of WHO Functional Class Change from Baseline Categorisation

| Planned Relative Time | WHO Category | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|
| Week 4 | n | XXX | XXX | XXX |
| | Improved | XX (%) | XX (%) | XX (%) |
| | No Change | XX (%) | XX (%) | XX (%) |
| | Deteriorated | XX (%) | XX (%) | XX (%) |
| | -2 | XX (%) | XX (%) | XX (%) |
| | -1 | XX (%) | XX (%) | XX (%) |
| | 0 | XX (%) | XX (%) | XX (%) |
| | +1 | XX (%) | XX (%) | XX (%) |
| | +2 | XX (%) | XX (%) | XX (%) |

Etc..

Note: Baseline is the last value recorded prior to start of study treatment

There are 4 grades of WHO FC based on symptom severity (Class I=none, Class IV=most severe).

Grades mapped to numeric scale 1-4 (i.e. Class IV=4).

Change categorisation (based on -2, -1, 0, +1, +2); No Change (0), Improved (-1,-2),

Deterioration (+1,+2).

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

Low dose, 2.5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ = 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

PPD

Programming notes: Present Weeks 4, 8, 12, 16, 20, 24 and EW, for each treatment group and overall.

Population: Intent-to-Treat

Table 2.12: Summary of plasma NT-Pro BNP concentration (ng/L)

| Treatment | Planned<br>Relative Time | n | Geometric<br>Mean | SD<br>[logs] | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Ambrisentan<br>Low Dose | Baseline* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | Week 12 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 24 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | EW | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Ambrisentan<br>High Dose | Baseline* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | Week 12 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 24 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | EW | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Total<br>(N=XXX) | Baseline*<br>Week 12<br>Week 24<br>EW | XXX<br>XXX<br>XXX | XX.X<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.XX<br>XX.XX | XX.X<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX<br>XX<br>XX | XX<br>XX<br>XX<br>XX |

Note:  $\star$  Baseline is the last value recorded prior to start of study treatment.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ =35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ =50 kg).

AMB112529

Protocol: AMB112529

Population: Intent-to-Treat

Table 2.14: Summary of Exploratory Echocardiogram

| Planned<br>Relative Time | | Ambrisentan<br>Low Dose | Ambrisentan<br>High Dose | Total |
|---|---|---|---|---|
| Baseline* | | (N=XXX) | (N=XXX) | (N=XXX) |
| Pericardial | N | XXX | XXX | XXX |
| Effusion | Absent | XX (%) | XX (%) | XX (%) |
| | Trace: separation of pericardial layers in both systole and diastole | XX (%) | XX (%) | XX (%) |
| | Small: diastolic separation equals 1cm | XX (%) | XX (%) | XX (%) |
| | Moderate: diastolic separation of 1 to 2cm | XX (%) | XX (%) | XX (%) |
| | Large: diastolic separation equals 2cm | XX (%) | XX (%) | XX (%) |
| Mean right | N | XXX | XXX | XXX |
| Atrial | Mean | XX.X | XX.X | XX.X |
| Pressure | SD | XX.XX | XX.XX | XX.XX |
| (mmHg) | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Tricuspid | N | XXX | XXX | XXX |
| Annular | Mean | XX.X | XX.X | XX.X |
| Plane | SD | XX.XX | XX.XX | XX.XX |
| Systolic | Q1 | XX.X | XX.X | XX.X |
| Excursion | Median | XX.X | XX.X | XX.X |
| (cm) | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion. EW = Early Withdrawal. Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ = 35 kg).

High dose, 5 mg (body weight >= 20 kg and < 35 kg); 7.5 mg (>= 35 kg and < 50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Present Baseline, Week 12, Week 24 and EW.

AMB112529

Protocol: AMB112529

Population: Intent-to-Treat

Table 2.14: Summary of Exploratory Echocardiogram

| Planned | | 7 | 7 1 | m - + - 1 |
|---|---|---|---|---|
| Relative Time | | Ambrisentan | Ambrisentan<br>High Dose | Total |
| Baseline* | | Low Dose<br>(N=XXX) | (N=XXX) | (N=XXX) |
| Dabetine | | (11 11111) | (11 212121) | (14 212121) |
| Eccentricity | N | XXX | XXX | XXX |
| Index | Mean | XX.X | XX.X | XX.X |
| Systolic | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Eccentricity | N | XXX | XXX | XXX |
| Index | Mean | XX.X | XX.X | XX.X |
| Diastolic | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

## PPD

Programming notes: Present Baseline, Week 12, Week 24 and EW.

Population: Intent-to-Treat

Protocol: AMB112529

Table 2.14: Summary of Exploratory Echocardiogram

| Planned<br>Relative Time | | Ambrisentan | Ambrisentan | Total |
|--------------------------|--------|-------------|-------------|---------|
| Relative lime | | Low Dose | High Dose | IOCAL |
| Baseline* | | (N=XXX) | (N=XXX) | (N=XXX) |
| Tricuspid | N | XXX | XXX | XXX |
| Regurgitant | Mean | XX.X | XX.X | XX.X |
| Jet Velocity | SD | XX.XX | XX.XX | XX.XX |
| (m/s) | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Right | N | XXX | XXX | XXX |
| Ventricular | Mean | XX.X | XX.X | XX.X |
| Pressure | SD | XX.XX | XX.XX | XX.XX |
| (mmHg) | Q1 | XX.X | XX.X | XX.X |
| . 3. | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

## PPD

Programming notes: Present Baseline, Week 12, Week 24 and EW.

Population: Intent-to-Treat

Protocol: AMB112529

Table 2.15: Summary of Change from Baseline in Exploratory Echocardiogram

| Pericardial n XXX XXX XXX Effusion No Change XX (%) | Planned | | | | |
|---|---|---|---|---|---|
| Week 12 (N=XXX) (N=XXX) (N=XXX) Pericardial n XXX (%) XXX (% | Relative Time | | Ambrisentan | Ambrisentan | Total |
| Pericardial n | | | Low Dose | High Dose | |
| Effusion No Change Absent Improved XX (%) | Week 12 | | (N=XXX) | (N=XXX) | (N=XXX) |
| Effusion No Change Absent Improved XX (%) | Pericardial | n | XXX | XXX | XXX |
| Absent XX (%) XX | Effusion | No Change | | | |
| Improved XX (%) | | | | | XX (%) |
| Mean right n XXX XXX XXX Atrial Mean XX.X XX.X XX.X Pressure SD XX.XX XX.XX XX.XX (mmHg) Q1 XX.X XX.X XX.X XX.X Q3 XX.X XX.X XX.X XX.X XX.X Min. XX XX XX XX Annular Mean XX.X XX.X XX.X Plane SD XX.XX XX.X XX.X XX.X Systolic Q1 XX.X XX.X XX.X XX.X Excursion Median XX.X XX.X XX.X XX.X XX.X (cm) Q3 XX.X XX.X XX.X XX.X XX.X XX.X Min. XX XX.X XX.X< | | Improved | | | XX (%) |
| Atrial Mean XX.X | | <del>-</del> | | | XX (%) |
| Atrial Mean XX.X | Mean right | n | XXX | XXX | XXX |
| (mmHg) Q1 XX.X | Atrial | Mean | XX.X | XX.X | XX.X |
| (mmHg) Q1 XX.X | Pressure | SD | XX.XX | XX.XX | XX.XX |
| Median XX.X | (mmHq) | | | | |
| Min. XX < | | Median | XX.X | XX.X | |
| Max. XX XX XX XX XXX | | Q3 | XX.X | XX.X | XX.X |
| Tricuspid n Annular Mean Plane SD Systolic Q1 Excursion Median (cm) Q3 Min. XXX XXX XXX XXX XX.XX XX.X | | Min. | XX | XX | XX |
| Annular Mean Plane SD Systolic Q1 Excursion Median (cm) Q3 Min. XX XX XX XX XX XX XX XX XX XX XX XX XX | | Max. | XX | XX | XX |
| Plane SD XX.XX XX | Tricuspid | n | XXX | XXX | XXX |
| Systolic Q1 Excursion Median (cm) Q3 Min. XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X | Annular | Mean | XX.X | XX.X | XX.X |
| Excursion Median XX.X XX.X XX.X (cm) Q3 XX.X XX.X XX.X Min. XX XX XX | Plane | SD | XX.XX | XX.XX | XX.XX |
| $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | Systolic | Q1 | XX.X | XX.X | XX.X |
| Min. XX XX XX | Excursion | Median | XX.X | XX.X | XX.X |
| | (cm) | Q3 | XX.X | XX.X | XX.X |
| Max. XX XX XX | | Min. | XX | XX | XX |
| | | Max. | XX | XX | XX |

Note: Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal. Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Programming notes: Present Week 12, Week 24 and EW.

Population: Intent-to-Treat

Table 2.15: Summary of Change from Baseline in Exploratory Echocardiogram

| Planned<br>Relative Time | | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|
| RCIGCIVE TIME | | Low Dose | High Dose | 10041 |
| Week 12 | | (N=XXX) | (N=XXX) | (N=XXX) |
| Eggentnigitu | | XXX | XXX | XXX |
| Eccentricity | n<br>Maar | | | |
| Index | Mean | XX.X | XX.X | XX.X |
| Systolic | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Eccentricity | N | XXX | XXX | XXX |
| Index | Mean | XX.X | XX.X | XX.X |
| Diastolic | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| | riax. | $\Lambda\Lambda$ | $\Lambda\Lambda$ | $\Lambda\Lambda$ |

Note: Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

## PPD

Programming notes: Present Week 12, Week 24 and EW.

Population: Intent-to-Treat

Table 2.15: Summary of Change from Baseline in Exploratory Echocardiogram

| Planned<br>Relative Time | | Ambrisentan | Ambrisentan | Total |
|--------------------------|--------|-------------|-------------|---------|
| | | Low Dose | High Dose | |
| Week 12 | | (N=XXX) | (N=XXX) | (N=XXX) |
| Tricuspid | N | XXX | XXX | XXX |
| Regurgitant | Mean | XX.X | XX.X | XX.X |
| Jet Velocity | SD | XX.XX | XX.XX | XX.XX |
| (m/s) | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Right | N | XXX | XXX | XXX |
| Ventricular | Mean | XX.X | XX.X | XX.X |
| Pressure | SD | XX.XX | XX.XX | XX.XX |
| (mmHg) | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

Note: Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

## PPD

Programming notes: Present Week 12, Week 24 and EW.

Population: Intent-to-Treat

Table 2.16: Summary of Cardiopulmonary Hemodynamics

| Parameter | Treatment | Planned<br>Relative Time | n | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| <parameter (units)=""></parameter> | Ambrisentan<br>Low Dose | Baseline* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | (N=XXX) | Week 24 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | EW | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Ambrisentan<br>High Dose | Baseline* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | (N=XXX) | Week 24 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | , | EW | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Total | Baseline* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | (N=XXX) | Week 24 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | , | EW | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |

Note:  $\star$  Baseline is the last value recorded prior to start of study treatment.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ =35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ =50 kg).

#### PPD

Programming notes: Include heart rate, mean arterial blood pressure, mean pulmonary arterial pressure, mean right atrial pressure, left ventricular end diastolic pressure or pulmonary capillary wedge pressure, pulmonary vascular resistance, cardiac output, cardiac index (calculated value), arterial oxygen saturation and mixed venous oxygen saturation.

Population: Intent-to-treat

Table 2.18: Summary of Number of Subjects with School Days within the Past Month

| Planned Relative Time Baseline* | Low Dose<br>(N=XX) | High Dose<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| Subjects with scheduled days Subjects with at least one scheduled day missed Number of scheduled days missed / Number of scheduled days | xx (xx%<br>xx (xx%<br>xx/xxx (xx% | ) xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx/xxx (xx%) |
| Subjects with at least one scheduled day missed due to PAH Number of scheduled days missed due to PAH / Number of scheduled days | xx (xx%<br>xx (xx%<br>xx/xxx (xx% | ) xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx/xxx (xx%) |

Note: \* Baseline is the last value recorded prior to start of study treatment.

This summary excludes subjects with 0 scheduled days of school for the given period.

There were no subjects with follow up visits (of the 3 subjects who did not participate in study AMB11488, one died, one was lost to follow-up and the other withdrew consent).

EW = Early Withdrawal.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Programming notes: Present Baseline, Weeks 4, 8, 12, 16, 20, 24 and EW.

Population: Intent-to-Treat

Table 2.19: Summary Statistics of School Days within the Past month

| | | | - 1 1 . | |
|-----------------------|--------|-------------|-------------|-------------|
| Planned Relative Time | | Ambrisentan | Ambrisentan | Total |
| D 1' # | | Low Dose | High Dose | /3T T77777\ |
| Baseline* | | (N=XXX) | (N=XXX) | (N=XXX) |
| Number | n | XXX | XXX | XXX |
| of scheduled days | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Number | N | XXX | XXX | XXX |
| of missed days | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Number | N | XXX | XXX | XXX |
| of missed days | Mean | XX.X | XX.X | XX.X |
| due to PAH | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

Note: \* Baseline is the last value recorded prior to start of study treatment.

This summary excludes subjects with 0 scheduled days of school for the given period.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal. Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >= 20 kg and < 35 kg); 7.5 mg (>= 35 kg and < 50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Present Baseline, Weeks 4, 8, 12, 16, 20, 24 and EW.

Population: Intent-to-Treat

Table 2.19: Summary Statistics of School Days within the Past month

| | | 7.1. | 7 1 1 | m |
|-----------------------|--------|---------------|-------------|---------|
| Planned Relative Time | | Ambrisentan | Ambrisentan | Total |
| | | Low Dose | High Dose | |
| Baseline* | | (N=XXX) | (N=XXX) | (N=XXX) |
| Proportion of days | n | XXX | XXX | XXX |
| missed (%) | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Proportion of days | N | XXX | XXX | XXX |
| missed due to PAH(%) | Mean | XX.X | XX.X | XX.X |
| ( ), | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX • X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX <b>.</b> X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| | ran. | XX | XX | ΛΛ |

Note: \* Baseline is the last value recorded prior to start of study treatment.

This summary excludes subjects with 0 scheduled days of school for the given period.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal. Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Programming notes: Present Baseline, Weeks 4, 8, 12, 16, 20, 24 and EW.
Population: Intent-to-Treat

Table 2.21: Summary of Subject Global Assessment (SF10 Health Survey for Children)

| Planned Relative Time | | Ambrisentan | Ambrisentan | Total |
|-------------------------|--------|-------------|-------------|---------|
| | | Low Dose | High Dose | |
| Baseline* | | (N=XXX) | (N=XXX) | (N=XXX) |
| Physical Health Summary | n | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Psychosocial Summary | N | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

PPD

Programming notes: Present Baseline, Weeks 4, 8, 12, 16, 20, 24 and EW.

Population: Intent-to-Treat

Table 2.23: Summary of SF10 Health Survey - Number and Percentage of Subjects with Particular Item Responses

| Planned Relative Time | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|
| | Low Dose | High Dose | |
| Baseline* | (N=XXX) | (N=XXX) | (N=XXX) |
| Completed SF-10 ^ | XX (%) | XX (%) | XX (%) |
| In general, would you say your child's health is | | | |
| n | XX | XX | XX |
| Excellent | XX (%) | XX (%) | XX (%) |
| Very Good | XX (%) | XX (%) | XX (%) |
| Good | XX (%) | XX (%) | XX (%) |
| Fair | XX (%) | XX (%) | XX (%) |
| Poor | XX (%) | XX (%) | XX (%) |
| During the past 4 weeks, has your child been limited doing | | | |
| things that take some energy such as riding a bike or skating | | | |
| due to HEALTH problems? | | | |
| n | XX | XX | XX |
| Yes, limited a lot | XX (%) | XX (%) | XX (%) |
| Yes, limited some | XX (%) | XX (%) | XX (%) |
| Yes, limited a little | XX (%) | XX (%) | XX (%) |
| No, not limited | XX (%) | XX (%) | XX (%) |
| During the past 4 weeks, has your child been limited during | | | |
| bending, lifting or stooping due to HEALTH problems? | | | |
| n | XX | XX | XX |
| Yes, limited a lot | XX (%) | XX (%) | XX (%) |
| Yes, limited some | XX (%) | XX (%) | XX (%) |
| Yes, limited a little | XX (%) | XX (%) | XX (%) |
| No, not limited | XX (%) | XX (%) | XX (%) |
| etc | | | |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion. EW = Early Withdrawal.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

#### PPD

Programming notes: Present Baseline, Weeks 4, 8, 12, 16, 20, 24 and EW.

<sup>^</sup> Completed at least one of the 10 items of SF-10

Table 3.1: Summary of Exposure to Investigational Product

| | | Ambrisentan | Ambrisentan | Total |
|------------------|---------------|-------------|-------------|---------|
| | | Low Dose | High Dose | |
| | | (N=XXX) | (N=XXX) | (N=XXX) |
| Number of days | n | XXX | XXX | XXX |
| of exposure | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Interval of days | n | XXX | XXX | XXX |
| of exposure | <=30 days | XX (%) | XX (%) | XX (%) |
| - | 31 to 60 days | XX (%) | XX (%) | XX (%) |
| | 61 to 90 days | XX (%) | XX (%) | XX (%) |
| | Etc | XX (%) | XX (%) | XX (%) |

Note: For each patient, exposure (days) = date of last dose of study drug - first dose date + 1 day. Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight >= 20 kg and <35 kg); 7.5 mg (>= 35 kg and <50 kg); 10 mg (>= 50 kg).

Table 3.2: Summary of Treatment-Emergent Adverse Events

| System Organ Class<br>Preferred term | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Any event | XX (%) | XX (%) | XX (%) |
| Gastrointestinal disorders | | | |
| Any event | XX (%) | XX (%) | XX (%) |
| Dyspepsia | XX (%) | XX (%) | XX (%) |
| Nausea | XX (%) | XX (%) | XX (%) |
| Nervous system disorders | | | |
| Any event | XX (%) | XX (%) | XX (%) |
| Headache | XX (%) | XX (%) | XX (%) |
| Dizziness | XX (%) | XX (%) | XX (%) |
| Somnolence | XX (%) | XX (%) | XX (%) |
| Tremor | XX (%) | XX (%) | XX (%) |
| Sedation | XX (%) | XX (%) | XX (%) |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Programming notes: Events will be sorted in descending order of total incidence across treatment groups for the System Organ Class and in descending order of total incidence for the preferred term within each System Organ Class. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Table 3.3: Summary of Treatment-Emergent Adverse Events by Preferred Term

| Preferred term | Ambrisentan<br>Low Dose<br>(N=XXX) | | Total<br>(N=XXX) |
|---|---|---|---|
| Any event | XX (%) | XX (%) | XX (%) |
| Dyspepsia | XX (%) | XX (%) | XX (%) |
| Nausea | XX (%) | XX (%) | XX (%) |
| Headache | XX (%) | XX (%) | XX (%) |
| Dizziness | XX (%) | XX (%) | XX (%) |
| Somnolence | XX (%) | XX (%) | XX (%) |
| Tremor | XX (%) | XX (%) | XX (%) |
| Sedation | XX (%) | XX (%) | XX (%) |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

### PPD

Programming notes: Events will be sorted in descending order of total incidence across treatment groups for the preferred term. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Table 3.4: Summary of Treatment-Emergent Adverse Events by Maximum Intensity

| | Ambrisentan Low Dose (N=XXX) | | | Ambrisentan High Dose (N=XXX) | | |
|---|---|---|---|---|---|---|
| | Mild | Moderate | Severe | Mild | Moderate | Severe |
| System Organ Class<br>Preferred Term | | | | | | |
| Any Event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Cardiovascular disorders | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Any Event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Hypertension | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Syncope | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Aneurysms | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Hypotension | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | | | | | | |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

# PPD

Programming notes: Repeat display for Total group on following page. Subjects who experience the same event several times, with different intensities/grades, will only be counted with the maximum intensity/grade. For example, a subject who had three headaches, two severe and one mild, is counted only once, under the preferred term "Headache" in the "Severe" column of the table. Likewise, each subject is counted only once, at the maximum severity/grade, within each SOC even though they may have several different PT events at different intensities/grades within that SOC. Events will be sorted in descending order of total incidence across treatment groups for the System Organ Class and in descending order of total incidence for the preferred term within each System Organ Class. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Table 3.5: Summary of Treatment-Emergent Adverse Events by Action Taken with IP

| System Organ Class<br>Preferred term<br>Action Taken | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Any event | XX (%) | XX (%) | XX (%) |
| <system 1="" class="" organ=""></system> | | | |
| <any event=""></any> | XX (%) | XX (%) | XX (%) |
| IP withdrawn | XX (%) | XX (%) | XX (%) |
| Dose interrupted | XX (%) | XX (%) | XX (%) |
| Dose reduced | XX (%) | XX (%) | XX (%) |
| Dose not changed | XX (%) | XX (%) | XX (%) |
| Dose increased | XX (%) | XX (%) | XX (%) |
| Not applicable | XX (%) | XX (%) | XX (%) |
| <preferred 1="" term=""></preferred> | XX (%) | XX (%) | XX (%) |
| IP withdrawn | XX (%) | XX (%) | XX (%) |
| Dose interrupted | XX (%) | XX (%) | XX (%) |
| Dose reduced | XX (%) | XX (%) | XX (%) |
| Dose not changed | XX (%) | XX (%) | XX (%) |
| Dose increased | XX (%) | XX (%) | XX (%) |
| Not applicable | XX (%) | XX (%) | XX (%) |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

# PPD

Programming notes: Subjects who experience the same event several times, with different Action Taken, will only be counted once for the overall and Preferred Term category, but more than once in the Action Taken categories. Events will be sorted in descending order of total incidence across treatment groups for the preferred term. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Population: Safety

Table 3.8: Summary of Cumulative Incidence of Treatment-Emergent Adverse Events by Time to First Occurrence

Treatment: Ambrisentan Low Dose (N=XXX)

| | | | Time S | Since Start | of Study | Medication | | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred term | <2 Wks | <4 Wks | <8 Wks | <12 Wks | <16 Wks | <20 Wks | <24 Wks | Overall |
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Gastrointestinal | | | | | | | | |
| disorders | | | | | | | | |
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dyspepsia | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Nausea | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Nervous system | | | | | | | | |
| disorders | | | | | | | | |
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Headache | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dizziness | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Somnolence | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Tremor | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Sedation | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

# PPD

Programming notes: Events will be sorted in descending order of total incidence across treatment groups for the preferred term. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order. Repeat for Ambrisentan High Dose and Total groups.

Table 3.10: Summary of Serious Treatment-Emergent Adverse Events - Number of Subjects and Occurrences

| System Organ Class<br>Preferred Term | Treatment<br>Group | Subjects<br>Affected,<br>Number | Subjects<br>Exposed,<br>Number | Occurrences<br>All, Number | Occurrences<br>Causally<br>Related to<br>Treatment,<br>Number* | Fatalities,<br>Number | Fatalities Causally Related to Treatment, Number* |
|---|---|---|---|---|---|---|---|
| CARDIAC DISORDERS | | | | | | | |
| Atrial fibrillation | Ambrisentan<br>Low Dose | | Х | х | X | X | Х |
| | Ambrisentan<br>High Dose | х | Х | х | X | Х | Х |
| | Total | X | Х | X | Х | X | X |
| Bradyarrhythmia | Ambrisentan<br>Low Dose | | Х | х | Х | X | Х |
| | Ambrisentan<br>High Dose | Х | Х | х | Х | X | Х |
| etc | Total | Х | X | Х | Х | х | х |

Note: \* Drug-related as determined by the investigator.

Table 3.11: Summary of Serious Treatment-Emergent Adverse Events by Outcome

| System Organ Class<br>Preferred term<br>Outcome | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Any event | XX (%) | XX (%) | XX (%) |
| <system 1="" class="" organ=""></system> | | | |
| <any event=""></any> | XX (%) | XX (%) | XX (%) |
| Recovered/Resolved | XX (%) | XX (%) | XX (%) |
| Recovering/Resolving | XX (%) | XX (%) | XX (%) |
| Recovered/Resolved with sequelae | XX (%) | XX (%) | XX (%) |
| Not Recovered/ Not Resolved | XX (%) | XX (%) | XX (%) |
| <preferred 1="" term=""></preferred> | XX (%) | XX (%) | XX (%) |
| Recovered/Resolved | XX (%) | XX (%) | XX (%) |
| Recovering/Resolving | XX (%) | XX (%) | XX (%) |
| Recovered/Resolved with sequelae | XX (%) | XX (%) | XX (%) |
| Not Recovered/ Not Resolved | XX (%) | XX (%) | XX (%) |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

# PPD

Programming notes: Subjects who experience the same event several times, with different Outcome, will only be counted once for the overall and Preferred Term category, but more than once in the Outcome categories. Events will be sorted in descending order of total incidence across treatment groups for the preferred term. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Table 3.21: Summary of Haematology Data

Parameter: <Parameter (units)>

| Treatment | Planned<br>Relative Time | N | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Ambrisentan | Baseline* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Low Dose | | | | | | | | | |
| (N=XXX) | Week 2 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 4 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 8 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 12 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 16 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 20 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 24 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | EW | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Ambrisentan<br>High Dose | Baseline* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | Week 2 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 4 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 8 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 12 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 16 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 20 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Week 24 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | EW | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Total<br>(N=XXX) | Etc | | | | | | | | |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up wisits. Of the 3 continuous start of the

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion. EW = Early Withdrawal. Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Table 3.23: Summary of Haematology Data of Potential Clinical Concern

Parameter: <Parameter (units) [Reference range = xx.x to xx.x]>

| Planned<br>Relative Time | Category | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|
| Baseline* | N | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 2 | N | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 4 | N | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 8 | N | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 12 | N | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion. EW = Early Withdrawal.

For 'Any time post-baseline':-

Subjects with both Normal and Low values are counted once under their worst case (Low).

Subjects with both Normal and High values are counted once under their worst case (High).

Subjects with both High and Low values are counted under both categories.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

Table 3.23: Summary of Haematology Data of Potential Clinical Concern

Parameter: <Parameter (units) [Reference range = xx.x to xx.x ]>

| Planned<br>Relative Time | Category | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|
| Week 16 | N | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 20 | N | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 24 | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| EW | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Any time post-baseline | n | XXX | XXX | XXX |
| _ | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

For 'Any time post-baseline':-

Subjects with both Normal and Low values are counted once under their worst case (Low).

Subjects with both Normal and High values are counted once under their worst case (High).

Subjects with both High and Low values are counted under both categories.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Table 3.29: Summary of Liver Events Assessment

| | | | High | Ambrisentan<br>High Dose<br>(N=XXX) | | Total (N=XXX) |
|---|---|---|---|---|---|---|
| Subjects reporting a significant liver chemistry result * Subjects with event occurring while receiving study treatment | XX<br>XX | (XX%)<br>(XX%) | XX<br>XX | (XX%)<br>(XX%) | XX<br>XX | (XX%)<br>(XX%) |
| Subjects with event occurring after stopping study treatment | XX | (XX%) | XX | (XX%) | XX | (XX%) |

Note: \* A significant liver chemistry result is any result which meets the stopping criteria defined in the protocol.

Detailed information on liver events assessment can be found in related listings.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Table 3.30 Summary of Vital Signs

| Parameter | Treatment | Planned<br>Relative Time | n | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| <parameter (units)=""></parameter> | Ambrisentan<br>Low Dose | Baseline* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | (N=XXX) | Week 2 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | , | Week 4 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 8 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 12 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 16 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 20 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 24 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | EW | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Ambrisentan<br>High Dose | Baseline* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | (N=XXX) | Week 2 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 4 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 8 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 12 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 16 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 20 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Week 24 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | EW | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Total<br>(N=XXX) | Etc | | | | | | | | |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal. Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

### PPD

Programming notes: Include Height, Weight, Systolic BP, Diastolic BP, Heart Rate, BSA and BMI.

Table 3.32: Summary of Vital Signs Data of Potential Clinical Concern

Parameter: <Parameter (units) [Reference range = xx.x to xx.x ]>

| Planned<br>Relative Time | Category | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|
| Baseline* | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 2 | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 4 | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 8 | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 12 | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

For 'Any time post-baseline':-

Subjects with both Normal and Low values are counted once under their worst case (Low).

Subjects with both Normal and High values are counted once under their worst case (High).

Subjects with both High and Low values are counted under both categories.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

PPD

Programming notes: Include Systolic BP, Diastolic BP and Heart Rate

Table 3.32: Summary of Vital Signs Data of Potential Clinical Concern

Parameter: <Parameter (units) [Reference range = xx.x to xx.x ]>

| Planned<br>Relative Time | Category | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|
| Week 16 | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 20 | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Week 24 | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| ΞW | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |
| Any time Post-baseline | n | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion.

EW = Early Withdrawal.

For 'Any time post-baseline':-

Subjects with both Normal and Low values are counted once under their worst case (Low).

Subjects with both Normal and High values are counted once under their worst case (High).

Subjects with both High and Low values are counted under both categories.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

PPD

Programming notes: Include Systolic BP, Diastolic BP and Heart Rate

Table 3.34: Summary of Physical Examination by Visit

| Planned Relative Time: Baseline | Low Dose<br>(N=XXX) | High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Ascites | | | |
| Absent | XX (%) | XX (%) | XX (%) |
| Present | XX (%) | XX (%) | XX (%) |
| Peripheral Oedema | | | |
| Absent | XX (%) | XX (%) | XX (%) |
| Present | XX (%) | XX (%) | XX (%) |
| Saturated Oxygen (units) | | | |
| N | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion. EW = Early Withdrawal.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >= 20 kg and <35 kg); 7.5 mg (>= 35 kg and <50 kg); 10 mg (>= 50 kg).

Table 3.34: Summary of Physical Examination by Visit

| Planned Relative Time: Week 12 | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|
| Ascites | | | |
| n | XX | XX | XX |
| Absent | XX (%) | XX (%) | XX (%) |
| Present: Improved | XX (%) | XX (%) | XX (%) |
| Present:Unchanged | XX (%) | XX (%) | XX (%) |
| Present:Worsened | XX (%) | XX (%) | XX (%) |
| Peripheral Oedema | | | |
| n | XX | XX | XX |
| Absent | XX (%) | XX (%) | XX (%) |
| Present: Improved | XX (%) | XX (%) | XX (%) |
| Abnormal:Worsened | XX (%) | XX (%) | XX (%) |
| Abnormal: Unchanged | XX (%) | XX (%) | XX (%) |
| Saturated Oxygen (units) | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not

participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion. EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight >= 20 kg and < 35 kg); 7.5 mg (>= 35 kg and < 50 kg); 10 mg (>= 50 kg).

#### PPD

Programming notes: Present for Week 12, Week 24 and EW.

Table 3.35: Summary of 12-lead ECG

| Planned<br>Relative Time | Category | Ambrisentan<br>Low Dose<br>(N=XXX) | Ambrisentan<br>High Dose<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|
| Baseline* | n | XXX | XXX | XXX |
| | Normal | XX (%) | XX (%) | XX (%) |
| | Abnormal, not clinically significant | XX (%) | XX (%) | XX (%) |
| | Abnormal, clinically significant | XX (%) | XX (%) | XX (%) |
| Week 12 | n | XXX | XXX | XXX |
| | Normal | XX (%) | XX (%) | XX (%) |
| | Abnormal, not clinically significant | XX (%) | XX (%) | XX (%) |
| | Abnormal, clinically significant | XX (%) | XX (%) | XX (%) |
| Week 24 | n | XXX | XXX | XXX |
| | Normal | XX (%) | XX (%) | XX (%) |
| | Abnormal, not clinically significant | XX (%) | XX (%) | XX (%) |
| | Abnormal, clinically significant | XX (%) | XX (%) | XX (%) |
| ΣW | n | XXX | XXX | XXX |
| | Normal | XX (%) | XX (%) | XX (%) |
| | Abnormal, not clinically significant | XX (%) | XX (%) | XX (%) |
| | Abnormal, clinically significant | XX (%) | XX (%) | XX (%) |
| Any time post-baseline | n | XXX | XXX | XXX |
| | Normal | XX (%) | XX (%) | XX (%) |
| | Abnormal, not clinically significant | XX (%) | XX (%) | XX (%) |
| | Abnormal, clinically significant | XX (%) | XX (%) | XX (%) |

Note: \* Baseline is the last value recorded prior to start of study treatment.

There were no subjects with post-last dose follow up visits. Of the 3 subjects who did not participate in study AMB115488, one died, one was lost to follow-up and the other was investigator discretion. EW = Early Withdrawal.

For 'Any time post-baseline' if a subject had more than one ECG result, the worst case will be chosen for a conservative approach.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

Table 3.36: Summary of Endocrinology assessments - Female

#### Overall

| Planned Relative Time | Ambrisentan | Ambrisentan | Total |
|-------------------------------|-------------|-------------|-----------|
| | Low Dose | High Dose | |
| Baseline* | (N=XXX) | (N=XXX) | (N=XXX) |
| Daseiine | (11-7/2/2) | (11-2222) | (11-2222) |
| Female breast development | | | |
| n | XXX | XXX | XXX |
| Pre-adolescent | XX (%) | XX (%) | XX (%) |
| Breast bud stage | XX (%) | XX (%) | XX (%) |
| Etc | XX (%) | XX (%) | XX (%) |
| Female pubic hair development | | | |
| n | XXX | XXX | XXX |
| Pre-adolescent | XX (%) | XX (%) | XX (%) |
| Sparse growth | XX (%) | XX (%) | XX (%) |
| Etc | XX (%) | XX (%) | XX (%) |

Note: \* Baseline is the last value recorded prior to start of study treatment.

EW = Early Withdrawal.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Pre-pubertal: Stage 1 breast development, Post-pubertal: Stage ≥ 2 breast development.

### PPD

Programming notes: Present for Baseline, Week 12, Week 24 and EW, Overall and by Pubertal Status (Pre-pubertal, Post Pubertal).

Table 3.37: Summary of Endocrinology assessments - Male Overall

| Planned Relative Time | Ambrisentan | Ambrisentan | Total |
|-------------------------|-------------|-------------|---------|
| | Low Dose | High Dose | |
| Baseline* | (N=XXX) | (N=XXX) | (N=XXX) |
| Right Testicular volume | | | |
| (units) | | | |
| N | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |
| Left Testicular volume | | | |
| (units) | | | |
| N | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |

Note:  $\star$  Baseline is the last value recorded prior to start of study treatment.  ${\tt EW}$  = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ =35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ = 50 kg).

Pre-pubertal: testicular volume < 4 ml, Post-pubertal: testicular volume ≥ 4 ml

# PPD

Programming notes: Present for Baseline, Week 12, Week 24 and EW, Overall and by Pubertal Status (Pre-pubertal, Post Pubertal).

Table 3.37: Summary of Endocrinology assessments - Male Overall

| Planned Relative Time | Ambrisentan<br>Low Dose | Ambrisentan<br>High Dose | Total |
|---|---|---|---|
| Baseline* | (N=XXX) | (N=XXX) | (N=XXX) |
| Male genital development | | | |
| N | XXX | XXX | XXX |
| Pre-adolescent | XX (%) | XX (%) | XX (%) |
| Etc | XX (%) | XX (%) | XX (%) |
| Male pubic hair development | | | |
| N | XXX | XXX | XXX |
| Pre-adolescent | XX (%) | XX (%) | XX (%) |
| Sparse growth | XX (%) | XX (%) | XX (%) |
| Etc. | XX (%) | XX (%) | XX (%) |

Note: \* Baseline is the last value recorded prior to start of study treatment.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Pre-pubertal: testicular volume < 4 ml, Post-pubertal: testicular volume ≥ 4 ml

# PPD

Programming notes: Present for Baseline, Week 12, Week 24 and EW, Overall and by Pubertal Status (Pre-pubertal, Post Pubertal).

Table 3.38: Summary of Pubertal Development Shifts from Baseline - Female Overall

Female Breast Development

| | Planned<br>Relative | Code | | Baseline Code | | | |
|---|---|---|---|---|---|---|---|
| Treatment | Time | | 1 | 2 | 3 | 4 | 5 |
| Ambrisentan Low Dose (N=XXX) | Week 12 | 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 3 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 4 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 5 | XX (%) | XX (%) | XX (%) | XX (%) | XX |
| | | Unknown/ | XX | XX | XX | XX | XX |
| | | Not Recorded | | | | | |
| | Week 24 | 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 3 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 4 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 5 | XX (%) | XX (%) | XX (%) | XX (%) | XX |
| | | Unknown/<br>Not Recorded | XX | XX | XX | XX | XX |

Etc..

Note: Baseline is the last value recorded prior to start of study treatment.

EW = Early Withdrawal.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ =35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ =50 kg).

Pre-pubertal: Stage 1 breast development, Post-pubertal: Stage  $\geq$  2 breast development.

# PPD

Programming notes: Present for Female Breast Development and Female Pubic Hair Development, for each treatment group, overall and by Pubertal Status (Pre-pubertal, Post Pubertal), at week 12, 24 and EW. Put coding below on first page on listing:-

Female Breast Development:-

1=Pre-adolescent; elevation of papilla only, 2=etc...

Female Pubic Hair Development:-

 $\mathbf{1}$ =Pre-adolescent; vellus over pubes not developed over anterior abdominal wall, 2=etc...

Table 3.39: Summary of Pubertal Development Shifts from Baseline - Male Overall

Male Genital Development

| | Planned<br>Relative | | | Baseline Code | | | |
|---|---|---|---|---|---|---|---|
| Treatment | Time | | 1 | 2 | 3 | 4 | 5 |
| Ambrisentan Low Dose (N=XXX) | Week 12 | 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 3 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 4 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 5 | XX (%) | XX (%) | XX (%) | XX (%) | XX |
| | | Unknown/ | XX | XX | XX | XX | XX |
| | | Not Recorded | | | | | |
| | Week 24 | 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 3 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 4 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 5 | XX (%) | XX (%) | XX (%) | XX (%) | XX |
| | | Unknown/<br>Not Recorded | XX | XX | XX | XX | XX |

Etc..

Note: Baseline is the last value recorded prior to start of study treatment.

EW = Early Withdrawal.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ =35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ =50 kg).

Pre-pubertal: testicular volume < 4 ml, Post-pubertal: testicular volume  $\geq$  4 ml

# PPD

Programming notes: Present for Male Genital Development and Male Pubic Hair Development, for each treatment group, overall and by Pubertal Status (Pre-pubertal, Post Pubertal), at week 12, 24 and EW. Put coding below on first page on listing:-

Male Genital Development:-

1=Pre-adolescent; testes, scrotum and penis same size and proportion, 2=etc...

Male Pubic Hair Development:-

 $\mathbf{1}$ =Pre-adolescent; velus over pubes no further developed than over abdominal wall, 2=etc...

Table 3.40: Summary of Testicular Volume Change from Baseline - Male Overall

| Planned Relative Time | | Ambrisentan | Ambrisentan | Total |
|-----------------------|--------|-------------|-------------|---------|
| | | Low Dose | High Dose | |
| | | (N=XXX) | (N=XXX) | (N=XXX) |
| Week 12 | N | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Week 24 | N | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Etc | | | | |

Note: Baseline is the last value recorded prior to start of study treatment.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

Pre-pubertal: testicular volume < 4 ml, Post-pubertal: testicular volume ≥ 4 ml

#### PPD

Programming notes: Present overall and by Pubertal Status (Pre-pubertal, Post Pubertal), at week 12, 24 and EW.

Population: Safety

Table 3.41: Summary of Change from Baseline in Plasma Endocrine Parameters - Female Overall

Parameter: <Parameter (units)>

| Planned Relative Time | | Ambrisentan<br>Low Dose | Ambrisentan<br>High Dose | Total |
|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) |
| Wools 12 | N | XXX | XXX | XXX |
| Week 12 | | | | |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Week 24 | N | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| E+ a | | | | |

Etc..

Note: Baseline is the last value recorded prior to start of study treatment.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ =35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ =50 kg).

Pre-pubertal: Stage 1 breast development, Post-pubertal: Stage ≥ 2 breast development.

#### PPD

Programming notes: Present overall and by Pubertal Status (Pre-pubertal, Post Pubertal), at week 12, 24 and EW, for Follicle Stimulating Hormone, Luteinizing Hormone, Sex Hormone Binding Globulin, Total Testosterone and Inhibin B.

Population: Safety

Table 3.41: Summary of Change from Baseline in Plasma Endocrine Parameters - Male Overall

Parameter: <Parameter (units)>

| Planned Relative Time | | Ambrisentan<br>Low Dose | Ambrisentan<br>High Dose | Total |
|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) |
| Week 12 | N | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Week 24 | N | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Etc | | | | |

Note: Baseline is the last value recorded prior to start of study treatment.

EW = Early Withdrawal.

Q1 = 1st quartile, Q3 = 3rd quartile.

Low dose, 2.5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

Pre-pubertal: testicular volume < 4 ml, Post-pubertal: testicular volume ≥ 4 ml

#### PPD

Programming notes: Present overall and by Pubertal Status (Pre-pubertal, Post Pubertal), at week 12, 24 and EW, for Follicle Stimulating Hormone, Luteinizing Hormone, Sex Hormone Binding Globulin, Total Testosterone and Inhibin B.


Protocol: AMB112529

Population: Intent-to-treat

Listing 1.1: Listing of Randomised and Actual Treatments

Country: Argentina
Centre ID: XXXXXX

| Centre<br>ID/<br>Subject<br>ID | Randomisation<br>Number / Date | Randomisation<br>Strata | Actual<br>Strata | Randomised /<br>Actual Treatment | Treatment<br>Start Date | Deviation [1] |
|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX / DDMMMYYYY | Aetiology - IPAH /<br>Age 12-18 | IPAH /<br>Age 12-18 | Low dose /<br>Low dose | DDMMMYYY | |
| XXXXXX | XXXXXX /<br>DDMMMYYYY | Aetiology - HPAH /<br>Age 12-18 | HPAH /<br>Age 12-18 | Low dose /<br>Low dose | DDMMMYYY | |

Note: 1 = Indicates subjects who have a deviation between their randomised and actual strata or treatment. IPAH, idiopathic PAH; HPAH, heritable [familial] PAH; PAH-CTD, secondary to connective tissue disease; PAH-CHD, persistent despite surgical repair of atrial/ventricular/atrio-ventricular septal defects, and persistent patent ductus.

Programming notes: Sort by Country, Centre ID, Subject ID.

Population: Intent-to-Treat

Listing 1.2: Listing of Reasons for Study Withdrawal

Treatment: Ambrisentan Low Dose

| Centre ID/ | Date of | Study | Reason for |
|------------|------------|-------|--------------|
| Subject ID | Withdrawal | Day | Withdrawal |
| XXXXXX/ | DDMMMYYYY | XX | XXXXXXXXXXXX |
| XXXXXX | | | |
| XXXXXX/ | DDMMMYYYY | XX | XXXXXXXXXXXX |
| XXXXXX | | | |
| XXXXXX/ | DDMMMYYYY | XX | XXXXXXXXXXXX |
| XXXXXX | | | |
| Etc | | | |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD


Protocol: AMB112529

Population: Intent-to-Treat

Listing 1.3: Listing of Subjects with Inclusion/Exclusion Criteria Deviations

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Туре | Criterion |
|---|---|---|
| XXXXXX/<br>XXXXXX | Inclusion | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | Exclusion | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD


Protocol: AMB112529

Population: Intent-to-Treat

Listing 1.4: Listing of Demographic Characteristics

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Partial<br>Date of Birth | Age (years)* | Sex | Child Bearing<br>Potential | Ethnicity |
|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | YYYY | XX | Female | Pre-menarcheal | Hispanic/Latino |

Etc..

Note: Age is based on full date of birth. Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD


Protocol: AMB112529

Population: Intent-to-Treat

Listing 1.5: Listing of Race

Treatment: Ambrisentan Low Dose

| Centre ID/ | |
|-------------------|-----------------------------|
| Subject ID | Race |
| XXXXXX/<br>XXXXXX | Asian - East Asian Heritage |
| Etc | |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Population: Intent-to-treat

# Listing 1.6: Listing of Disease History

Treatment: Ambrisentan Low Dose

| Centre ID /<br>Subject ID | Diagnosis | Sub category | Date of<br>Diagnosis | Duration<br>of PAH<br>(yrs) | Baseline<br>WHO FC |
|---|---|---|---|---|---|
| XXXXXX /<br>XXXXXX | Idiopathic PAH | | DDMMMYYYY | Х.Х | I |
| XXXXXX /<br>XXXXXX | Persistent PAH despite surgical repair | Atrio-ventricular septal defects | DDMMMYYYY | X.X | II |
| Etc | | | | | |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD


Protocol: AMB112529

Population: Intent-to-Treat

Listing 1.7: Listing of Medical Conditions

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Age (y)/<br>Sex/ | Classification | Preferred Term | Condition | Status |
|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX | Hepatobiliary disorders | xxxxxxxxxxxx | HEPATITIS A | Current |
| | | Psychiatric disorders | XXXXXXXXXXXXXX | PARANOIA COMBINED WITH MANIA. | Past |
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX | Eye disorders | XXXXXXXXXXXXXXX | ASTIGMATISM | Current |
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX | Metabolism and nutrition disorders | XXXXXXXXXX | RICKETS | Current |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Etc..

Population: Intent-to-Treat

Listing 1.8: Listing of Medications

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | | Unit<br>Dose/ | | |
|---|---|---|---|---|
| | ATC Level 1/ | Units/ | Date | Date |
| | Ingredient/ | Freq/ | Started/ | Stopped/ |
| | Verbatim Text | Route | Study Day | Study Day |
| | | | | _ |
| XXXXXX/ | Endocrine & metabolic/ | 2/ | PPD | |
| XXXXXX | Fluticasone propionate/ | MG/ | 15 | |
| | FLIXOTIDE # | 2XD/ | | |
| | | IH | | |
| | Endogrino ( motabolio/ | 4 / | PPD | Ongoing |
| | Endocrine & metabolic/ | - / | | Ongoing |
| | Fluticasone propionate/ | MG/ | 21 | |
| | FLIXOTIDE # | 2XD/ | | |
| | | IH | | |

Etc..

Etc..

Note: \* Prior, # Concomitant, \$ Post-treatment.

PAH Therapies are not included within this listing, for PAH Therapy please see Listing 1.7 Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD
Population: Intent-to-Treat

Listing 1.9: Listing of PAH Therapy

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Drug Class/<br>ATC Level 1/<br>Ingredient/<br>Verbatim Text/ | Total<br>Daily<br>Dose/<br>Units | Date<br>Started/<br>Study Day | Date<br>Stopped/<br>Study Day | Reason the medication discontinued or changed? |
|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | X/<br>XX | DDMMMYYYY/<br>XX | DDMMMYYYY | XXXXXXXXXXXXX |
| XXXXXX/<br>XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | X/<br>XX | DDMMMYYYY/<br>XX | Ongoing | XXXXXXXXXXXX |

Etc..

Etc..

Note: \* Prior, # Concomitant, \$ Post-treatment.
@ Ongoing background PAH therapy at baseline
Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).
High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.

Population: Intent-to-Treat

Listing 1.10: Relationship between ATC Level 1, Ingredient and Verbatim Text

| ATC Level 1 | Ingredient | Verbatim Text |
|---|---|---|
| Endocrine & metabolic | Fluticasone Propionate<br>Prednisolone | FLIXOTIDE<br>PREDNISOLONE |
| Drugs acting via the nervous system | Paracetamol | PANADOL<br>CHILDREN'S PANADOL 1-5YERS |
| Etc | | |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Sort by ATC level 1treatment group, Ingredient.

AMB112529

Protocol: AMB112529

Population: Intent-to-Treat

Listing 1.11: Listing of Protocol Deviation

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Important<br>Protocol<br>Deviations | Protocol Deviation Category | Protocol Deviation<br>Description | Protocol<br>Deviation<br>Date/<br>Study Day | Visit Phase | Action taken |
|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | Y | Biological specimen sample procedures | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>XX | XXXXXXX | XXXXXXXXXX<br>XXXXXXXXXX<br>X |
| XXXXXX/<br>XXXXXX | N | Other: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>XX | xxxxxxx | XXXXXXXXXX<br>XXXXXXXXXX<br>X |

Etc..

Etc..

Note: \* Important Deviation

Low dose, 2.5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ = 35 kg).

High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

PPD

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.


Protocol: AMB112529

Population: Intent-to-Treat

Listing 2.1: Listing of 6 Minute Walk Distance Data

Treatment: Ambrisentan Low Dose

| Centre ID/ | | | Dis | stance Walked | l (m) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Visit | Visit<br>Date/<br>Study Day | Actual | Change<br>from<br>Baseline | Percentage<br>Change<br>from<br>Baseline | Did subject walk less than 6 minutes?/ Reason for stopping prematurely | Duration<br>walked<br>(seconds) | Did subject<br>use<br>supplemental<br>oxygen | Oxygen<br>flow<br>rate<br>(L/min) |
| XXXXXX/<br>XXXXXX | XXXXXXX | DDMMMYYYY/<br>XX | XXX | | | Y/<br>XXXXXXXXXXXX | XXX | Y | XXXX |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXX | XXX | XXX | Y/<br>XXXXXXXXXXXX | XXX | Y | XXXX |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXX | XXX | XXX | N | | N | |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXX | XXX | XXX | N | | N | |
| | Etc | | | | | | | | |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

### PPD


Protocol: AMB112529

Population: Intent-to-Treat

Listing 2.2: Listing of Clinical Worsening of PAH

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Event Date/<br>Study Day | Clinical worsening criteria |
|---|---|---|
| XXXXXX/ | DDMMMYYYY/ | Hospitalisation for worsening of PAH |
| XXXXXX | XX<br>DDMMMYYYY/<br>XX | PAH related deterioration: Clinical signs or symptoms of right sided heart failure |
| Etc | 7777 | |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.

Population: Intent-to-Treat

Listing 2.3: Listing of WHO Functional Class Data

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Visit | Visit<br>Date/<br>Study Day | WHO pulmonary hypertension functional classification | Actual<br>* | Change<br>from<br>Baseline | Change<br>Categorisation |
|---|---|---|---|---|---|---|
| XXXXXX/ | XXXXXXX | DDMMMYYYY/ | Class II | 2 | | |
| XXXXXX | XXXXXXX | XX<br>DDMMMYYYY/<br>XX | Class II | 2 | 0 | NC |
| | XXXXXXX | DDMMMYYYY/<br>XX | Class IV | 4 | 2 | Det |
| | XXXXXXX | DDMMMYYYY/<br>XX | Class I | 1 | -1 | Imp |
| | Etc | | | | | |

Etc..

Note: There are 4 grades for WHO FC based on severity of symptoms (Class I = none, Class IV = most severe).

\* Grades mapped to numeric scale 1-4 (i.e. Class IV = 4).

Change categorisation (based on -2, -1, 0, +1, +2); NC=No Change (0), Imp=Improved (-1,-2),

Det=Deterioration (+1,+2).

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Population: Intent-to-Treat

Listing 2.4: Listing of Plasma NT-Pro BNP Concentration (ng/L)

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Visit | Visit<br>Date/<br>Study Day | Visit | t Value | Change from Baseline | |
|---|---|---|---|---|---|---|
| | | | Raw | Log | Raw | Log* |
| XXXXXX/<br>XXXXXX | XXXXXXX | DDMMMYYYY/<br>XX | XXX.X | X.XX | | |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXX.X | X.XX | XXX.X | X.XX |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXX.X | X.XX | XXX.X | X.XX |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXX.X | X.XX | XXX.X | X.XX |
| | Etc | | | | | |

Etc..

Note: \* Log (change from baseline) = Log (Visit) - Log (Baseline). Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

# PPD


Protocol: AMB112529

Population: Intent-to-Treat

Listing 2.5: Listing of Exploratory Echocardiogram

Treatment: Ambrisentan Low Dose

| Centre<br>ID/<br>Subject<br>ID | Visit | Visit<br>Date/<br>Study Day | Pericardial<br>effusion/<br>Change from<br>Baseline | Mean right atrial pressure (mmHg)/Change from Baseline | Tricuspid annular plane systolic excursion (cm)/ Change from Baseline | Systolic<br>Eccentricity<br>Index/<br>Change from<br>Baseline | Diastolic<br>Eccentricity<br>Index/<br>Change from<br>Baseline | Tricuspid<br>regurgitant<br>jet (m/s)/<br>Change from<br>Baseline | Right Ventricular Pressure (mmHg)/ Change from Baseline |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX/ | XXXXXXX | DDMMMYYYY/ | Absent | XXX | XXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXXXXXX | XX<br>DDMMMYYYY/<br>XX | Trace/<br>Worsened | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX |
| | XXXXXXX | DDMMMYYYY/<br>XX | Small/<br>Worsened | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX |
| | XXXXXXX | DDMMMYYYY/ | Trace/ | XXX/ | XXX/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | Etc | XX | Worsened | XXX | XXX | XXX | XXX | XXX | XXX |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

### PPD


Protocol: AMB112529

Population: Intent-to-Treat

Listing 2.6: Listing of Cardiopulmonary Hemodynamics

Treatment: Ambrisentan Low Dose

| Centre ID/ | | | | Mean Pulmonary | Mean Right | Pulmonary |
|---|---|---|---|---|---|---|
| Subject ID | | Right Heart | Heart | Arterial | Atrial | Capillary Wedge |
| | | Catheterization | Rate(bpm)/ | Pressure (mmHg)/ | Pressure (mmHg)/ | Pressure (mmHg)/ |
| | | Date / | Change from | Change from | Change from | Change from |
| | Visit | Study Day | Baseline | Baseline | Baseline | Baseline |
| XXXXXX/ | XXXXXXX | DDMMMYYYY/ | XXX | XXX | XXX | XXX |
| XXXXXX | | XX | | | | |
| | XXXXXXX | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | | XX | XXX | XXX | XXX | XXX |
| | XXXXXXX | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | | XX | XXX | XXX | XXX | XXX |
| | XXXXXXX | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | | XX | XXX | XXX | XXX | XXX |
| | Etc | | | | | |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Population: Intent-to-Treat

Listing 2.6: Listing of Cardiopulmonary Hemodynamics

Treatment: Ambrisentan Low Dose

| Visit | Right Heart<br>Catheterization<br>Date /<br>Study Day | Method used to Calculate Cardiac Output/Oxygen Consumption | Cardiac Output<br>(Litres/minute)/<br>Change from<br>Baseline | Cardiac index (L/min/meters/ square)/ Change from Baseline | Pulmonary Vascular<br>Resistance<br>(mmHg/L/min)/<br>Change from<br>Baseline |
|---|---|---|---|---|---|
| XXXXXXX | DDMMMYYYY/<br>HH:MM/ | XXXXXXXXXXX/<br>XXXXXXXXXXX | XXX | XXX | XXX |
| XXXXXXX | DDMMMYYYY/<br>HH:MM/ | XXXXXXXXXXX/<br>XXXXXXXXXXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX |
| XXXXXXX | DDMMMYYYY/<br>HH:MM/ | XXXXXXXXXXX/<br>XXXXXXXXXXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX |
| XXXXXXX | DDMMMYYYY/<br>HH:MM/<br>XX | XXXXXXXXXXXX/<br>XXXXXXXXXXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX |
| | xxxxxx<br>xxxxxx | Catheterization Date / Visit Study Day XXXXXXX DDMMMYYYY/ HH:MM/ XX XXXXXXX DDMMMYYYY/ HH:MM/ XX XXXXXXX DDMMMYYYY/ HH:MM/ XX XXXXXXX DDMMMYYYY/ HH:MM/ XX XXXXXXX DDMMMYYYY/ HH:MM/ XX | Right Heart Calculate Catheterization Date / Oxygen Visit Study Day Consumption XXXXXXX DDMMMYYYY/ XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Right Heart Cardiac Output/ (Litres/minute)/ Date / Oxygen Change from Baseline XXXXXXX DDMMMYYYY/ XXXXXXXXXXXX XXX XXX XXXXXXX DDMMMYYYY/ XXXXXXXXXXX XXX XXX XXXXXX DDMMMYYYY/ XXXXXXXXXXX XXX XXX XXX XXX XXX XXXXXX | Right Heart Calculate Cardiac Output (L/min/meters/ Catheterization Cardiac Output/ (Litres/minute)/ square)/ Date / Oxygen Change from Change from Study Day Consumption Baseline Baseline XXXXXXX DDMMMYYYY/ XXXXXXXXXXXX XXX HH:MM/ XXXXXXXXXXXX XXX XXX XXX XXXXXXX DDMMMYYYY/ XXXXXXXXXXX XXX XXX XXX XXXXXXX DDMMMYYYY/ XXXXXXXXXXX XXX XXX XXX XXX XXX |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

### PPD

Population: Intent-to-Treat

Listing 2.6: Listing of Cardiopulmonary Hemodynamics

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Visit | Right Heart<br>Catheterization<br>Date /<br>Study Day | Left Ventricle<br>End Diastolic<br>Pressure (mmHg)/<br>Change from<br>Baseline | Arterial Oxygen Saturation Percentage/ Change from Baseline | Venous<br>Oxygen<br>Saturation/<br>Change from<br>Baseline | Mean Arterial<br>Pressure (mmHg)/<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|
| XXXXXX/ | XXXXXXX | DDMMMYYYY/ | XXX | XXX | XXX | XXX |
| XXXXXX | | HH:MM/ | ****** | 212121 | 71717 | 22222 |
| | XXXXXXX | XX<br>DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | XXXXXXX | HH:MM/ | XXX | XXX | XXX | XXX |
| | XXXXXXX | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | | HH:MM/<br>XX | XXX | XXX | XXX | XXX |
| | XXXXXXX | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | | HH:MM/<br>XX | XXX | XXX | XXX | XXX |
| | Etc | | | | | |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Population: Intent-to-Treat

Listing 2.7: Listing of School Days

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Age(y)/<br>Sex/<br>Race | Visit | Visit Date /<br>Study Day | School Days<br>Scheduled */<br>Change from<br>Baseline | School Days<br>missed/<br>Change from<br>Baseline | School Days<br>missed due<br>to PAH/<br>Change from<br>Baseline | Proportion of days missed (%)/ Change from Baseline | Proportion of days missed due to PAH (%)/Change from Baseline |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/<br>Male/ | Baseline | DDMMMYYYY/<br>XX | XX | XX | XX | XX | XX |
| XXXXX | XXXXXX | XXXXXXX | DDMMMYYYY/<br>XX | XX/<br>XX | XX/<br>XX | XX/<br>XX | XX/<br>XX | XX/<br>XX |
| | | XXXXXXX | DDMMMYYYY/<br>XX | XX/<br>XX | XX/<br>XX | XX/<br>XX | XX/<br>XX | XX/<br>XX |
| | | XXXXXX | DDMMMYYYY/<br>XX | XX/<br>XX | XX/<br>XX | XX/<br>XX | XX/<br>XX | XX/<br>XX |

Etc..

Etc..

Note: \* In past month at Baseline; since baseline visit at Week 4; and since the patient's last clinic visit (all other assessments).

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Population: Intent-to-Treat

Listing 2.8: Listing of Subject Global Assessment (SF10 Health Survey for Children)

Treatment: Ambrisentan Low Dose

Centre ID/ Subject ID

| | Visit | Visit Date<br>/<br>Study Day | 1.Childs<br>General<br>Health | 2a.Limited<br>Riding and<br>Skating | 2b.Limited<br>Bending | 3.Physical<br>Problems<br>Limit<br>Schoolwork | 4.Emotional<br>Problems<br>Limit<br>Schoolwork | 5.Bodily pain |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/ | XXXXXXX | DDMMMYYYY/ | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |
| XXXXXX | XXXXXXX | XX<br>DDMMMYYYY/ | XXXXXXX | XXXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |
| | 17171717171717 | XX | ************ | ************ | 1717171717171717 | 1717171717171717 | 1717171717171717 | */*/*/*/*/*/ |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |
| | Etc | 2323 | | | | | | |

Etc..

Note: The Physical Summary Score (aggregate of item responses 1, 2a, 2b, 3 and 5) and Psychosocial Summary Score (aggregate of item responses 4, 6, 7, 8 and 9) were calculated by QualityMetrics Health Outcomes software.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Population: Intent-to-Treat

Listing 2.8: Listing of Subject Global Assessment (SF10 Health Survey for Children)

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Visit | Visit Date<br>/<br>Study Day | 6.Satisfied with friendships | 7.Satisfied with life overall | 8.Time<br>bothered or<br>upset | 9.General<br>behaviour | Physical<br>Health<br>Summary/<br>Change<br>from<br>Baseline | Psychosocial<br>Summary/<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/ | XXXXXXX | DDMMMYYYY/ | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XX/ | XX/ |
| XXXXXX | | XX | | | | | XX | XX |
| | XXXXXXX | DDMMMYYYY/ | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XX/ | XX/ |
| | | XX | | | | | XX | XX |
| | XXXXXXX | DDMMMYYYY/ | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XX/ | XX/ |
| | | XX | | | | | XX | XX |
| | XXXXXXX | DDMMMYYYY/ | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XX/ | XX/ |
| | | XX | | | | | XX | XX |
| | Etc | | | | | | | |

Etc..

Note: The Physical Summary Score (aggregate of item responses 1, 2a, 2b, 3 and 5) and Psychosocial Summary Score (aggregate of item responses 4, 6, 7, 8 and 9) were calculated by QualityMetrics Health Outcomes software.

Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Listing 3.1: Listing of Exposure and Compliance to Investigational Product

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | IP<br>Start<br>Date | IP<br>Stop<br>Date | Duration<br>(Days) | % of<br>compliant<br>visits | Visit | Visit Date/<br>Study Day | Compliance since the last visit |
|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | DDMMMYYYY | DDMMMYYYY | XX | 100 | XXXXXXXX | DDMMMYYYY/<br>XX | |
| 77777777 | | | | | XXXXXXXX | DDMMMYYYY/<br>XX | >=80% and <=120% |
| | | | | | XXXXXXXX | DDMMMYYYY/<br>XX | >=80% and <=120% |

Etc..

Note: Compliant visits are those at which subjects are >=80% and <=120% compliant. Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Listing 3.2: Listing of All Adverse Events

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Age (y)/<br>Sex/<br>Race/<br>Weight (kg) | Preferred Term/<br>Verbatim Text | Outcome/<br>Onset Date/<br>Resolution<br>Date/<br>Frequency | Time Since<br>First Dose/<br>Last Dose/<br>Duration (days) | Maximum<br>Intensity/<br>Serious/<br>Withdrawal | Action<br>Taken/<br>Relation to<br>Study Drug |
|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX/<br>XXXXXX/<br>XX | XXXXXXXXXX/<br>XXXXXXXXXX *<br>XXXXXXXXXX/<br>XXXXXXXXXX | XXXXXXXX/ DDMMMYYYY/ DDMMMYYYY/ XXXXXXXXX XXXXXXXX/ DDMMMYYYY/ DDMMMYYYY/ XXXXXXXXX | XX/<br>XX/<br>XX<br>XX/<br>XX/<br>XX/ | XXXX/<br>XXX/<br>XXX<br>XXXX/<br>XXX/<br>XXX | XXXXXXX/<br>XX<br>XXXXXXXX/<br>XX |
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX/<br>XXXXXX/<br>XX | XXXXXXXXXX/<br>XXXXXXXXXXX \$ | XXXXXXXX/<br>DDMMMYYYY/<br>DDMMMYYYY/<br>XXXXXXXXX | XX/<br>XX/<br>XX | XXXX/<br>XXX/<br>XXX | XXXXXXXX/<br>XX |

Etc..

Note: \* Prior, # Treatment-emergent, \$ Post-treatment. Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID and Onset date.

Population: Safety

Listing 3.3: Listing of Relationship between Adverse Event System Organ Class, Preferred Term and Verbatim Text

| System Order Class | Preferred Term | Verbatim Text |
|---|---|---|
| Blood and lymphatic system disorder | Lymphadenopathy | Enlarged lymph node |
| Cardiac disorder | Palpitations<br>Tachycardia nos | Heart palpitation<br>Tachycardia |
| Etc | | |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Continue for all combinations. Sort in order of SOC, PT, and verbatim text.

Page 1 of n Population: Safety

Listing 3.4: Listing of Subject Numbers for Specified Adverse Events

Treatment: Ambrisentan Low Dose

| System Organ Class | No. with | Centre ID/Subject ID |
|---|---|---|
| Preferred term | Event | |
| Gastrointestinal disorders | | |
| Dyspepsia | 9 | XXXXXX/XXXXXX, XXXXXX/XXXXXX, XXXXXX/XXXXXX, XXXXXX/XXXXXX, XXXXXX/XXXXXX, XXXXXX/XXXXXX, XXXXXX/XXXXXX, |
| Nausea<br>Etc | 1 | XXXXXX/XXXXXX |

Note: Low dose, 2.5 mg (body weight  $\geq$ =20 kg and  $\leq$ 35 kg); 5 mg ( $\geq$ = 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>=50 kg).

PPD

Programming notes: Present each treatment group. Sort by treatment group, SOC, PT.

Listing 3.8: Listing of Haematology

Central Laboratory

Treatment: Ambrisentan Low Dose

| Centre ID/ | Age(y)/ | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Sex/ | | | | | | | | | |
| | Race/ | | Planned | | | | | | | |
| | Baseline | | Relative | | Study | Converte | ed Data | Fla | ag ' | ξ |
| | Weight(kg) | Lab test (units) | Time | Date | Day | Value | Normal Range | NR | CC | BL |
| XXXXXX/<br>XXXXXX | XX/ | <parameter (units)=""></parameter> | Screening | DDMMMYYYY | XX | XXX | XXX - XXX | | | |
| | XXXXXX/ | | Baseline | DDMMMYYYY | XX | XXX | XXX - XXX | | | |
| | XXXXXX/ | | Week 2 | DDMMMYYYY | XX | XXX | XXX - XXX | Н | Н | Н |
| | XX | | Week 4 | DDMMMYYYY | XX | XXX | XXX - XXX | Н | | Н |
| | | | Week 8 | DDMMMYYYY | XX | XXX | XXX - XXX | | | |
| | | | Week 12 | DDMMMYYYY | XX | XXX | XXX - XXX | | | |
| | | | Week 16 | DDMMMYYYY | XX | XXX | XXX - XXX | | | |
| | | | Week 20 | DDMMMYYYY | XX | XXX | XXX - XXX | L | L | L |
| | | | EW | DDMMMYYYY | XX | XXX | XXX - XXX | | | |
| | | | Follow-Up | DDMMMYYYY | XX | XXX | XXX - XXX | L | | |

<Parameter (units)> Etc..

Etc..

Note: \* NR for Normal Range flag, CC for Clinical Concern flag; BL for Change from Baseline H=Above range, L=Below range
Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).
High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

### PPD

Listing 3.9 Listing of Haematology Data for Subjects with Abnormalities of Potential Clinical Concern

Central Laboratory

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Age(y)/<br>Sex/<br>Race/<br>Baseline | | | Planned<br>Relative | | Study | y Converted Data | | | | Fl | Flag * | * |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Weight(kg) | Lab test | (units) | Time | Date | Day | Value | Normal<br>Range | Low<br>Concern | High<br>Concern | NR | CC | BL |
| XXXXXX/<br>XXXXXX | XX/ | <paramete< th=""><th>er (units)&gt;</th><th>Screening</th><th>DDMMMYYYY</th><th>XX</th><th>XXX</th><th>XXX - XXX</th><th>XXX</th><th>XXX</th><th></th><th></th><th></th></paramete<> | er (units)> | Screening | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | XXXXXX/ | | | Baseline | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | XXXXXX/ | | | Week 2 | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | Н | Н | Н |
| | XX | | | Week 4 | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | Н | | Н |
| | | | | Week 8 | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | | | | Week 12 | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | | | | Week 16 | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | | | | Week 20 | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | L | L | L |
| | | | | EW | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | | | | Follow-Up | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | L | | |

<Parameter (units)> Etc..

Etc..

Note: \* NR for Normal Range flag, CC for Clinical Concern flag; BL for Change from Baseline H=Above range, L=Below range
Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).
High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

### PPD


Protocol: AMB112529
Population: Safety

Listing 3.13: Listing of Liver Event Results and Time of Event Relative to Treatment

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Age (y)/<br>Sex/<br>Race/ | Event Date/<br>Study Day | Days from<br>first dose to<br>start of<br>event | Days from<br>last dose to<br>start of<br>event | Event that reached or exceeded protocol defined criteria |
|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/ | DDMMMYYYY/ | X | X | ALT (alanine aminotransferase) |
| | XXXXXX/<br>XXXXXX/<br>XX | XX | | | |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.

Listing 3.14: Listing of patient specific information for liver events

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Age<br>(y)/<br>Sex/<br>Race/ | Event that reached or exceeded protocol defined criteria | Event<br>Date/<br>Study Day | Days from last dose to start of | Assessment | Result |
|---|---|---|---|---|---|---|
| XXXXXX/ | XX/ | XXXXXXXXXXXX | <u> </u> | | Subject become pregnant? | No |
| XXXXXX | XXXXXX/<br>XXXXXX/<br>XX | | XX | | Was a biopsy taken? Any unconventional medications Fasting or significant dietary change Is this event serious? Evaluation interval | Yes No No Yes During the treatment period |
| | | | | | Does the subject consume alcohol? Average number of units of alcohol consumed per week | Yes<br>XX |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.

Listing 3.15: Listing of Medical Conditions for Subjects with Liver Events on Treatment

| Treatment | Centre<br>ID/<br>Subject<br>ID | Age (y)/<br>Sex/<br>Race/ | Classification | Condition | Status |
|---|---|---|---|---|---|
| Ambrisentan<br>Low Dose | XXXXXX/<br>XXXXXX | XX/<br>XXXXXXX/<br>XXXXXX | Hepatobiliary | HEPATITIS A | Current |
| | | | Psychiatric | PARANOIA COMBINED WITH MANIA. | Past |
| | XXXXXX/<br>XXXXXX | XX/<br>XXXXXXX/<br>XXXXXX | Eye | ASTIGMATISM | Current |
| Ambrisentan<br>High Dose | XXXXXX/<br>XXXXXX | XX/<br>XXXXXXX/<br>XXXXXX | Metabolism and nutrition | RICKETS | Current |


Protocol: AMB112529
Population: Safety

Listing 3.16: Listing of Liver Biopsy Details

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Age<br>(y)/<br>Sex/ | Event that reached or exceeded protocol defined | Biopsy<br>Date/ | Biopsy<br>Size | | |
|---|---|---|---|---|---|---|
| | Race/ | criteria | Study Day | (mm) | Liver biopsy test | Liver biopsy result |
| XXXXXX/<br>XXXXXX | XX/ | XXXXXXXXXXXX | DDMMMYYYY/ | X | Bile ducts | Other: Bile ducts blocked |
| | XXXXXX/<br>XXXXXX/ | | XX | | Final diagnosis Description of liver cells/hepatocytes | Alcoholic hepatic cirrhosis<br>Normal |
| | XX | | | | Liver cell/hepatocyte inclusion/vacuole | No inclusions |
| | | | | | <pre>Hepatocyte/liver cell nuclear abnorm Etc</pre> | None |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.


Protocol: AMB112529
Population: Safety

Listing 3.17: Listing of Liver Imaging Details

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Age<br>(y)/<br>Sex/<br>Race/ | Event that reached or exceeded protocol defined criteria | Imaging<br>Date/<br>Study Day | Liver<br>imaging<br>method | Are images<br>technically<br>adequate? | | imaging test | Liver imaging result |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/ | XXXXXXXXXXXX | DDMMMYYYY/ | X | XX | Liver | Size | Hypertrophy (or enlarged) |
| AAAAAA | XXXXXX/<br>XXXXXX/ | | XX | | | Liver | Texture | Normal Not applicable - No |
| | 7171717171 | | | | | Liver | fatty infiltrate grade | fatty infiltration |
| | XX | | | | | Ascite | es present | None present<br>Not applicable - no |
| | | | | | | Gallst<br>Bilia | hepatic lesions character cones or gallbladder lesions by ductal lesions l/Hepatic vein abnormalities | hepatic lesions None None None |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.

Listing 3.18: Listing of Vital Signs

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Age(y)/<br>Sex/<br>Race | Visit | Visit<br>Date/<br>Study Day | Systolic Blood Pressure (mmHg)/ Change from Baseline | Diastolic Blood Pressure (mmHg)/ Change from Baseline | Heart Rate (bpm)/ Change from Baseline | Height (units)/ Change from Baseline | Weight (units)/ Change from Baseline | BMI<br>(units)/<br>Change<br>from<br>Baseline | BSA (units)/<br>Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX/<br>XXXXXX | XXXXXXX<br>XXXXXXX | DDMMMYYYY/ XX DDMMMYYYY/ XX DDMMMYYYY/ XX | XX/ XX/ XX XX/ XXX | XX<br>XX/<br>XX<br>XX/<br>XX | XX/ XX/ XX XX/ XX | XX/ XX/ XX XX/ XX | XX/ XX/ XX XX/ XX | XX/ XX/ XX XX/ XX | XX<br>XX/<br>XX<br>XX/<br>XX |

Etc..

Etc..

Note: H=Above clinical concern, L=Below clinical concern, Change from Baseline HC=Above clinical concern, LC=Below clinical concern Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg).

High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD


Protocol: AMB112529
Population: Safety

Listing 3.20: Listing of Physical Examination

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | Age(y)/<br>Sex/<br>Race | Visit | Visit<br>Date/<br>Study Day | Liver<br>Size | Jugular<br>Venous<br>Pressure | Ascites | Peripheral<br>Oedema | Saturated<br>Oxygen<br>(units) |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX/ | XXXXXXX | DDMMMYYYY/<br>XX | XXXXXX | XXXXXXX | XXXXXX | XXXXXXX | XX.XXX |
| *************************************** | XXXXXX | XXXXXXX | DDMMMYYYY/<br>XX | XXXXXX | XXXXXXXX (I) | XXXXXXX | XXXXXXX | XX.XXX |
| | | XXXXXXX | DDMMMYYYY/<br>XX | XXXXXX | XXXXXXX | XXXXXXX (W) | XXXXXX | XX.XXX |
| | | XXXXXXX | DDMMMYYYY/<br>XX | XXXXXX | XXXXXXXX (U) | XXXXXXX | XXXXXX | XX.XXX |

Etc..

Note: I=Improved, W=Worsened, U=Unchanged Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

# PPD


Protocol: AMB112529
Population: Safety

Listing 3.21: Listing of 12-Lead ECG Findings

Treatment: Ambrisentan Low Dose

| Centre ID/ | | | | |
|------------|---------|---------|-------------|--------------|
| Subject ID | Age(y)/ | | | |
| | Sex/ | | Visit Date/ | |
| | Race | Visit | Study Day | Result |
| XXXXXX/ | XX/ | XXXXXXX | DDMMMYYYY/ | XXXXXXXXXXXX |
| XXXXXX | XXXXXX/ | | XX | |
| | XXXXXX | XXXXXXX | DDMMMYYYY/ | XXXXXXXXXXXX |
| | | | XX | |
| | | XXXXXXX | DDMMMYYYY/ | XXXXXXXXXXXX |
| | | | XX | |
| | | Etc | | |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Listing 3.22: Listing of Endocrinology Assessments

Treatment: Ambrisentan Low Dose

| XXXXXXX | Centre ID/<br>Subject ID | Age(y)/<br>Sex/<br>Race | Visit | Endocrinology<br>Assessment<br>Date/<br>Study Day | Assessment Type | Assessment<br>Result |
|---|---|---|---|---|---|---|
| XXXXXXX Male genital XXXXXXXXX development XXX Male pubic hair XXXXXXXXX development XXX X | · | XX/ | | DDMMMYYYY/ | Testicular volume | _ |
| XX Right/Left (units) Male genital XXXXXXXXXX development XXX Male pubic hair XXXXXXXXX development XXX Etc XXXXXXX DDMMMYYYY/ Female breast XXXXXXXXXX XXXXXXX Female/ XXXXXXX Female/ XXXXXXXX Etc Etc | AAAAA | | | AA | Male genital<br>development<br>Male pubic hair | XXX<br>XXXXXXXXX |
| Male pubic hair XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | XXXXXXX | • | Right/Left (units)<br>Male genital | XXXXXXXXX |
| XXXXXX/ XX/ XXXXXXX DDMMMYYYY/ Female breast XXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXX | | | Et C | | Male pubic hair | |
| XXXXXXX Female/ XX development XXX Female pubic hair XXXXXXXXXX development XXX Etc | | | | | | |
| | • | Female/ | XXXXXXX | · | development<br>Female pubic hair | XXX<br>XXXXXXXXX |
| | E+ - | | Etc | | | |

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>=35 kg). High dose, 5 mg (body weight  $\geq$ 20 kg and  $\leq$ 35 kg); 7.5 mg ( $\geq$ 35 kg and  $\leq$ 50 kg); 10 mg ( $\geq$ 50 kg).

#### PPD


Protocol: AMB112529 Population: Safety

Listing 3.23: Listing of Pregnancy Results

Treatment: Ambrisentan Low Dose

| Centre ID/<br>Subject ID | | | | | |
|---|---|---|---|---|---|
| | Age(y)/ | | Visit Date/ | | Subject became |
| | Race | Visit | Study Day | Result | pregnant? |
| | | | | | _ |
| XXXXXX/ | XX/ | XXXXXXX | DDMMMYYYY/ | XXXXXXXXXXXX | No |
| XXXXXX | XXXXXX/ | | XX | | |
| | XXXXXX | XXXXXXX | DDMMMYYYY/ | XXXXXXXXXXXX | |
| | | | XX | | |
| | | XXXXXXX | DDMMMYYYY/ | XXXXXXXXXXXX | |
| | | | XX | | |
| | | Etc | | | |

Etc..

Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

#### PPD

Population: Intent-to-Treat

Protocol: AMB112529

Figure 1.1: Summary of Subject Accrual



Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Change Labels: X -> Ambrisentan Low Dose, Y -> Ambrisentan High Dose.

Figure 3.1: Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to First Treatment-Emergent Adverse Event



Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Programming notes: Change Labels: Drug A -> Ambrisentan Low Dose, Drug B -> Ambrisentan High Dose. Also present combined group. Annotate to display number of events in each group also.

Protocol: AMB112529
Population: Safety

Figure 3.3: Bar Chart of Treatment-Emergent Adverse Events Occurring in Two or More Subjects in any Treatment Group



Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Programming notes: Change Labels: DrugA -> Ambrisentan Low Dose, DrugB -> Ambrisentan High Dose. Also present combined group. Continue for each preferred term.

Figure 3.4: Box plots of Haematology Data by Week (Selected Parameters)

Parameter = <Parameter (units)>



Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

# PPD

Programming notes: Change Labels: Drug A -> Ambrisentan Low Dose, Drug B -> Ambrisentan High Dose. Also present combined group. Label vertical axes with parameter name and units. Label horizontal axis with appropriate week structure. Repeat for each parameter. Haematology parameters (haemoglobin, hematocrit, platelets), Chemistry parameters (Total bilirubin, AST, ALT, GGT, Creatinine). Use log scale for Plasma NT-Pro BNP (Figure 2.6 and Figure 2.7).

Figure 3.8: Patient Profiles of Liver Function Tests



Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

## PPD

Programming notes: Change Labels: Drug A -> Ambrisentan Low Dose, Drug B -> Ambrisentan High Dose. Also present combined group. Present parameters ALT, AST, Alk. Phos, Total Bilirubin. Present one patient per page only, not grid of 4 patients.

Figure 3.11: Line plots of Endocrinology Assessments by Subject



Note: Low dose, 2.5 mg (body weight >=20 kg and <35 kg); 5 mg (>= 35 kg). High dose, 5 mg (body weight >=20 kg and <35 kg); 7.5 mg (>=35 kg and <50 kg); 10 mg (>= 50 kg).

PPD

Programming notes: Only one patient on a page, with a grid of plots on each page for each parameter. For Figure 3.11, plot female breast development and pubic hair development; male testicular volume, genital development and pubic hair development and change from baseline in male testicular volume (left and right separately). For Figure 2.8 (Japanese subset) plot echocardiogram parameters. For coded data, plot the numeric code and present codes on first page of the plot.

# 19. APPENDICES

# 19.1. Appendix 1 – IDSL Age Calculation

IDSL standard/GSK standard of the derivation of AGE:

```
AGE = intck('year',DEMO.BIRTHDT, AGEREFDT) -

(month(AGEREFDT) < month(DEMO.BIRTHDT) or

(month(AGEREFDT)=month(DEMO.BIRTHDT) and

day(AGEREFDT) < day(DEMO.BIRTHDT)

));
```

For this study, it was decided that the AGE is calculated based on the date of the baseline visit ie.

AGEREFDT = Date of record with VISITNUM=20 in the VISIT dataset.

BIRTHDT = derived by DM in DEMO dataset which contains imputed date for date of birth (ie. 30JUNYYYY).